# SELFIe-HF

# PATIENT <u>SELF</u>-MANAGEMENT WITH HEMODYNAM<u>I</u>C MONITORING: VIRTUAL HEART FAILURE CLINIC AND OUTCOMES

A preliminary study in high risk patients Protocol Number: MHICC-2018-001

<u>Principal Investigator</u> Anique Ducharme, M.D., M.Sc.

Montreal Heart Institute 5000 Belanger Street (S-2700)

Montreal, Quebec, H1T 1C8 Phone: (514) 376-3330 ext. 3947

Fax: (514) 593-2575

<u>Co-Investigators</u>

Jean L. Rouleau, M.D. Anita Asgar, M.D., M.Sc. Jocelyn Dupuis, M.D., Ph.D. Simon de Denus, B. Pharm, PhD Montreal Heart Institute 5000 Belanger Street

Montreal, Quebec, H1T 1C8 Phone: (514) 593-7431

#### **Coordinating Center**

Montreal Health Innovations Coordinating Center 4100 Molson Street, Suite 400 Montreal (Quebec), H1Y 3N1

#### Project Leader

Hélène Brown, RN, B.Sc. CCRP Montreal Heart Institute

Phone: (514) 376-3330 ext. 3931

Fax: (514) 593-2575

#### An investigator initiated study

Montreal Heart Institute

This protocol contains information that is confidential and proprietary of Dr. Anique Ducharme and the Montreal Heart Institute

Protocol No: MHICC-2018-001

Version: FINAL 10

### DATE OF PROTOCOL: 01-JUN-2020

# **Signature Approval Page**

By signing below, I indicate that I have reviewed the Clinical Protocol in its entirety and approve its contents.

| Signature: | | Date: |
|---|---|---|
| | Dr. Anique Ducharme, MD<br>Principal Investigator<br>MHI | |
| Signature: | | Date: |
| | Marie-Claude Guertin, PhD<br>Lead Biostatistics<br>MHICC | |
| Signature: | | Date: |
| | Ourida Mehenni Hadjeres, MD<br>Lead Medical and Safety<br>MHICC | |
| Signature: | | Date: |
| | Andreas Orfanos, MBBCh, FFPM, MBA<br>Director<br>MHICC | |


## INVESTIGATOR'S STATEMENT AND SIGNATURE

| Protocol Title: Patient <u>SELF</u> -management with hemodynam <u>I</u> c monitoring: Virtual <u>H</u> eart <u>F</u> ailure Clinic and Outcomes. A preliminary study in high risk patients |
|---|
| Protocol Number: Version 10 |
| Version Date: 01-JUNE-2020 |
| I have read the protocol and agree to conduct this trial in accordance with all stipulations of the protocol, with applicable laws and regulations and in accordance with the ethical principles outlined in the Declaration of Helsinki. |
| By signing below, I hereby declare that I am not debarred, disqualified, or otherwise restricted by any agency from conducting any research studies. |
| Site Principal Investigator: |
| Signature: Date: |
| Printed Name: Anique Ducharme |
| Site Name: Montreal Heart Institute |

Protocol No: MHICC-2018-001 Version: FINAL 10

# Synopsis

| Title | Patient' <u>SELF</u> -management with HemodynamIc monitoring: virtual <u>Heart</u> |
|---|---|
| | <u>Failure clinic and outcomes (the SELFIe-HF trial): program.</u> |
| Investigator | CardioMEMS <sup>TM</sup> HF System |
| Device | |
| Study objectives | To demonstrate that a virtual Heart Failure Clinic (HFC) based on patient self-management using Pulmonary Artery Pressure (PAP) monitoring is superior to usual care of HFC, leads to decreased: hospital admissions for heart failure (HF), emergency department consultation and/or unplanned intravenous heart failure therapy and cardiovascular death, compared to a regular HFC, has low device-related complications and is cost-effective, in New York Heart Association (NYHA) class III and II (requiring diuretics) patients. |
| Study design | This will be a single center, prospective, randomized, open-label blinded-endpoint (PROBE) trial in which the treatment group will be implanted with a CardioMEMS HF sensor and managed using remote access to hemodynamics compared to a non-implanted control group. Patients with at least one hospitalization for HF (≥1) in the previous year (12 months) will be randomized into two groups, regardless of LVEF: ■ Usual care with the specialized multidisciplinary HF clinic team (Non-implanted Control) or ■ Hemodynamic monitoring, less intense HF clinic follow-up, and remote follow-up by a nurse clinician and patient empowerment with access to the PAP data (CardioMEMS group). Primary and secondary endpoints will be compared between groups after 12 months of follow-up and within groups comparing baseline parameters with 12 month follow-up measurements. |
| <b>Key Inclusion</b> | 1. Male or female ≥ 18 years old |
| criteria | <ol> <li>Symptomatic HF (NYHA III) with recent heart failure admission in the previous year (12 months). or</li> <li>Patient with at least one ER visit or unplanned HF clinic requiring iv diuretics within 12 months will be eligible if they have in addition a N-terminal pro-BNP (NT-proBNP) level &gt; 800pg/ml at screening AND NYHA Class II on diuretics (furosemide ≥ 40mg qd), III or ambulatory IV.</li> <li>HF with reduced or preserved EF of at least 3 months duration.</li> <li>Minimum technological knowledge either with a smartphone or iPAD for use of the self-management application, including access to internet.</li> </ol> |

#### 6 Anatomical criteria

- a. PA branch diameter between 7 mm 15 mm
- b. For BMI >35, distance from patient's back to the target PA<10 cm.

# **Key exclusion** criteria

- 1. Recent cardiovascular events: Acute coronary syndrome, percutaneous coronary intervention (PCI), new cardiac rhythm management (CRM) device (pacemaker, implantable cardioverter defibrillator (ICD) and cardiac resynchronization therapy (CRT)), CRM system revision, lead extraction or cardiac or other major surgery or transient ischemic attack or stroke within 2 months (3 months for CRT or cardiac surgery).
- 2. Scheduled cardiac surgery;
- 3. History of pulmonary embolism or recurrent deep vein thrombosis
- 4. Persistent NYHA Class IV and American College of Cardiology (ACC)/ American Heart Association (AHA) HF Stage D, patients implanted with a ventricular assist device (VAD), or patients listed for cardiac transplantation and likely to be transplanted within 12 months
- 5. Coexisting severe obstructive valvular lesions, obstructive hypertrophic cardiomyopathy, endocarditis, tamponade or large pericardial effusion
- 6. Clinically too unstable to be followed remotely; this includes but is not limited to:
  - a) Resting systolic blood pressure < 80 or > 180 mmHg;
  - b) Resting heart rate > 100 bpm;
  - c) Stage IV or V chronic kidney disease (Estimated Glomerular Filtration Rate (eGFR) that remains < 30mL/min/1.73m<sup>2</sup> by MDRD) or nonresponsive to diuretic therapy or on chronic renal dialysis;
- 7. Severe pulmonary hypertension with systolic pulmonary artery pressure ≥ 80 mmHg.
- 8. Pulmonary hypertension other than group II PH;
- 9. Anemia requiring transfusions, iron infusions, or hemoglobin below 100;
- 10. Coagulopathy or uninterruptible anticoagulation therapy or contraindication to antiplatelet/anticoagulant treatments anticipated in the protocol;
- 11. Intolerance to aspirin or clopidogrel;
- 12. Active infection requiring systemic antibiotics;
- 13. Life expectancy <1 year;

| Primary | The primary endpoint is the time to first occurrence of any component of |
|---|---|
| Endpoint | The primary endpoint is the time to first occurrence of any component of |
| Enupoint | the composite event as adjudicated by the Clinical Event Committee |
| | (CEC). Components of the event are: acute decompensated heart failure |
| | requiring emergency department consultation and/or unplanned |
| | intravenous heart failure therapy in an outpatient clinic, or hospital |
| | admission for heart failure or cardiovascular (CV) death during 12 months |
| | of follow-up. |
| Secondary | • |
| Endpoints primary endpoint | |
| • | • Changes from baseline in functional ability: |
| | NYHA class |
| | <ul> <li>Health-related Quality of life, as measured by a HF-specific</li> </ul> |
| | instrument (KCCQ) |
| | o 6-minute walk distance |
| | • Cost-effectiveness |
| | Device related endpoints |
| | <ul> <li>Safety: adverse events related to the device</li> </ul> |
| | <ul> <li>Number of successful patient contacts (virtual and clinic)</li> </ul> |
| | <ul> <li>PA pressures: changes, frequency of elevated readings</li> </ul> |
| | <ul> <li>Ease of application utilization.</li> </ul> |
| Tertiary/ | Goal for best practice |
| Exploratory | <ul> <li>% achieved target dose of guidelines derived medical therapy</li> </ul> |
| endpoints | (GDMT) (HF with reduced ejection fraction (HFrEF)) |
| | <ul> <li>Medication changes (mean dose achieved by class)</li> </ul> |
| | o Time (days) to achieve target doses of GDMT (HFrEF) |
| | Changes in cardiac remodeling assessed by echocardiography between |
| | baseline and 12 months: |
| | o indexed LV End-systolic and end-diastolic volumes (LVESVi, |
| | LVEDVi), left ventricular ejection fraction (LVEF) |
| | o Right ventricle (RV) dimensions and function, |
| | <ul> <li>Left atrium volume</li> </ul> |
| | <ul> <li>mitral and tricuspid regurgitation severity</li> </ul> |
| | Changes in specific biomarkers for heart failure |
| | Arrhythmia burden |
| | • Patient quality of life and satisfaction regarding both the virtual follow- |
| | up itself & the personalized algorithm using the application. |
| | Sample for drug concentrations |
| Control Group | Eligible patients who agreed to participate and provide informed consent |
| | that are randomly assigned to the control group will be followed using |
| | standard clinical management at the Montreal Heart Institute specialized |
| | HF clinic. |

Protocol No: MHICC-2018-001 Version: FINAL 10

| CardioMEMS<br>Group | Eligible patients who provide informed consent and randomized to the intervention group will be implanted with the CardioMEMS HF System and instructed to use the Patient Electronic System. In addition, patients will be provided the MyCardioMEMS smartphone app, which will include PA pressure information and instructions for any changes in therapy. |
|---|---|
| Number of subjects | 150 patients with 1:1 randomization |
| Plan for | For the primary endpoint, the analysis will be an unadjusted comparison of |
| statistical | time to first event. Event-rate curves will be estimated by the Kaplan-Meier |
| analysis | product-limit method and the difference between groups will be assessed |
| | using the log-rank test. Components of the primary endpoint will be |
| | analyzed similarly. |
| | ANCOVA models will be used to compare the secondary endpoints |
| | expressed as a change from baseline to 12 months between groups. The |
| | models will include fixed effects for group and baseline value as a |
| | covariate. Difference between groups in other continuous endpoints will be |
| | tested by either two-sample t-tests or Wilcoxon rank-sum tests depending |
| | on the distribution of the data. Chi-square tests will be used for categorical |
| | endpoints. |
| | All statistical tests will be two-sided and conducted at the 0.05 significance |
| | level. Statistical analysis will be done using SAS version 9.4 or higher. |

#### List of abbreviations

ACC American College of Cardiology ACE Angiotensin Converting Enzyme ADHF Acute Decompensated Heart Failure

AE Adverse Event AF Atrial Fibrillation

AHA American Heart Association
ARO Academic Research Organization

BMI Body Mass Index BPM Beat Per Minute

BNP B-type Natriuretic Peptide

BP Blood Pressure
BSA Blood Surface Area
BUN Blood Urea Nitrogen
CBC Complete Blood Count

CCTN Canadian Cardiac Transplantation Network

CEC Clinical Event Committee

CardioMEMS Heart sensor Allows Monitoring of Pulmonary Pressures

CHAMPION Heart Failure Patients Trial CHF Chronic Heart Failure

COPD Chronic Obstructive Pulmonary Disease

CRF Case Report Form

CRM Cardiac Rythm Management

CRT Cardiac Resynchronization Therapy

CV Cardiovascular

DCC Data Coordinating Center

DSMB Data and Safety Monitoring Board

ECG Electrocardiogram

eGFR estimated Glomerular Filtration Rate

ED Emergency Department EF Ejection Fraction

ePAD estimated Pulmonary Artery Diastolic

ER Emergency Room

ERA Endothelin Receptor Antagonist FDA Food and Drug Administration

GCP Good Clinical Practice

GDMT Guidelines Derived Medical Therapy

H Hour

HF Heart Failure

HFC Heart Failure Clinic

HfpEF Heart Failure with preserved Ejection Fraction
HfrEF Heart Failure with reduced Ejection Fraction
HFDMP Heart Failure Disease Management Program


HR Heart Rate

hs-CRP high-sensitivity C-Reactive Protein
ICD Implantable Cardioverter Defibrillator
ICER Incremental Cost- Effectiveness Ratio

IEC Independent Ethic Committee
IHM Implanted Hemodynamic Monitor

IRB Institutional Review Board

LA Left Atrium

LAP Left Atrial Pressure

LV Left ventricle

LVEF Left Ventricular Ejection Fraction

LVESi Left Ventricular volume indexed to BSA MDRD Modification of Diet in Renal Disease

Mg Milligram
Min Minute
mL Milliliter

mmHg millimeters of mercury

Mmol Millimol

MHI Montreal Heart Institute

MHICC Montreal Health Innovations Coordinating Center

MLHF Minnesota Living With Heart Failure
MRA Mineralocorticoid Receptor Antagonists

NT-proBNP N-terminal prohormone B-type Natriuretic Peptide

NYHA New York Heart Association

PA Pulmonary Artery

PAP Pulmonary Artery Pressure

PCI Percutaneous Coronary Intevention PCWP Pulmonary Capillary Wedge Pressure

PDE5I Phosphodiesterase 5 Inhibitors PH Pulmonary Hypertension

PIIINP Procollagen type III N-terminal Propeptide

pg/ml Picogram per millilter

PROBE Prospective Randomized Open-label Blinded-Endpoint

PVR Pulmonary Vascular Resistance
QALY Quality Adjusted Life Year
Qd quaque die (every day)

QOL Quality Of Life

RHC Right Heart Catherization

RV Right Ventricle

SAE Serious Adverse Event

SGCS Solube guynylate cyclase stimulators

SID Subject identification number VAD Ventricular Assist Device

VT/VF Ventricular Tachycardia/Ventricular Fibrillation

WHO World Health Organization


## **Table of Contents**

| List of | abbreviations | 8 |
|---|---|---|
| Table o | of Contents | 10 |
| 1. | RATIONALE | 12 |
| 1.1 | Background | 12 |
| 2. | Hypothesis: | 16 |
| 2.1 | Primary Hypothesis | 16 |
| 3. | STUDY OBJECTIVES | 17 |
| 4.1 | Primary Endpoint | 17 |
| 4.2 | Secondary Endpoints | 17 |
| 4.2.1 | Time to the first occurrence of the individual components of the composite endpoint | 17 |
| 4.2.2 | Changes in functional capacity between baseline and 12-months | 17 |
| 4.2.3 | Device-related endpoints (for intervention group only) | 17 |
| 4.2.4 | Cost-effectiveness | 18 |
| 4.3 | Tertiary/Exploratory Endpoints | 19 |
| 4.3.1 | Goal for best practice | 19 |
| 4.3.2 | Changes in echocardiographic parameters between baseline and 12 months | 19 |
| 4.3.3 | Changes in biomarkers levels between baseline and 12-months | 19 |
| 4.3.4 | Arrhythmia Burden | 19 |
| 4.3.5 | Patient quality of life and satisfaction | 19 |
| 4.3.6 | Drugs concentration | 19 |
| 5. | STUDY PROTOCOL | 20 |
| 5.1 | Study design | 20 |
| 5.2 | Inclusion/Exclusion Criteria | 21 |
| 5.2.1 | Inclusion Criteria | 21 |
| 5.2.2 | Exclusion Criteria | 22 |
| 5.3 | Subject Attribution Number | 23 |
| 6. | SUBJECT EVALUATION | 24 |
| 6.1 | Informed Consent | 24 |
| 6.2 | Visits 24 | |
| 7. | FLOW CHART | 28 |

| 8. SAI | -ETY | 29 |
|---|---|---|
| 8.1.<br>Event | Definition of Adverse Events, Serious Adverse Events, and procedures for reporting Serious Advers | |
| 8.1.1. | Adverse Event (AE) | 33 |
| 8.1.2. | Serious Adverse Event definition(SAE) | 33 |
| 8.1.6. | Procedures for Adverse Event reporting | 34 |
| 8.1.6.1 | . Investigator Reporting | 34 |
| 9. | STATISTICAL ANALYSIS | 35 |
| 9.1. | Sample size | 36 |
| 10. | INVESTIGATOR'S REGULATORY OBLIGATIONS | 36 |
| 10.1. | Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approval | 36 |
| 10.2. | Informed Consent | 37 |
| 10.3. | Declaration of Helsinki | 37 |
| 10.4. | Case Report Form | 37 |
| 10.5. | Confidentiality | 37 |
| 11. | DATA QUALITY ASSURANCE | 38 |
| 11.1. | Monitoring, Audits and inspections | 38 |
| 11.2. | Archiving | 39 |
| 12. | DATA MANAGEMENT | 39 |
| 13. | TRIAL COMMITTEES | 39 |
| 13.1. | Clinical Events Committee | 39 |
| 13.2. | Data and Safety Monitoring Board (DSMB) | 40 |
| Propos | ed Table 1. Patient Characteristics at Enrollment | 41 |
| Propos | ed Table 2. Changes in the main Parameters between baseline and 12-months in Survivors | 43 |
| Propos | ed Table 3. Pharmacological Profiles and Goal for best practice at 12 months | 44 |
| Propos | ed Table 4: Device related endpoints | 45 |
| Appen | dix 1: Elevated PA Mean Pressure – General Treatment Strategies in Protocol | 53 |
| Appen<br>financi | dix 2: Hospital admissions at Montreal Heart Institute with a primary diagnosis of heart failure, al year April 1st 2016 to March 31st 2017 | 54 |
| Appen | dix 3: Example of an individualized therapeutic plan | 55 |
| Appen | dix 4 World Medical Association Declaration of Helsinki | 56 |

#### 1.0 RATIONALE

#### 1.1 Background

Heart failure (HF) represents a major public health concern and its incidence will continue to rise as the population ages. The growing burden of HF on healthcare costs is well documented. Despite major advances in diagnosis and treatment, HF is associated with high rates of decompensation, hospitalization and mortality. Developing new approaches for patients with HF are essential. In the past, major efforts have been directed toward reducing length of stay by the development of performance measures, with the intent to improve post-discharge outcomes. Recently, however, the focus has shifted towards 30-day post-discharge readmission rates as a measure of quality of care due to important changes in reimbursement patterns in the US.

Congestion is one of the hallmarks of HF hospitalizations and an increase in body weight seems to be associated with HF-related hospitalizations, usually beginning at least one week before admission for acutely decompensated heart failure (ADHF).<sup>4</sup> Consequently, increased daily weight may identify a high risk period during which one can intervene to avert ADHF requiring hospitalization.<sup>5</sup>

In addition to congestion, the presence of pulmonary hypertension (PH) secondary to heart failure, classified as World Health Organization (WHO) Group 2 PH<sup>6</sup> is associated with increased morbidity and mortality.<sup>7</sup> Therefore, in theory, an elevated pulmonary artery pressure (PAP) and increased pulmonary vascular resistance (PVR) should represent meaningful triggers for therapeutic interventions, and the reduction of decompensated HF an attractive therapeutic target. HF management programs which rely on patients' empowerment through education and careful follow-up, as well as pharmacological and device-optimization have been shown to decrease hospital admissions, emergency consultations, improve quality of life and probably survival.<sup>8</sup> Unfortunately, due to resource limitations and the increasing number of patients with moderate to severe heart failure, the majority of patients that could benefit from follow-up in multidisciplinary heart failure clinics (HFC) do not readily have access to them in a timely manner.<sup>9</sup> Innovative approaches might be crucial to changing the emphasis of the HFC and processes. New transitional models for HF care have been developed, such as structured telephone care (or telehealth) with


symptoms and vital signs monitoring, home visits, use of technology and remote monitoring systems to reduce HF-related hospitalizations, but with mixed results.<sup>10-12</sup> Recently, the BEAT-HF trial failed to show a benefit for 30 and 180 days readmission or mortality using a combined approach of health coaching telephone calls and telemonitoring with electronic equipment for daily information (BP, HR, symptoms and weight);<sup>13</sup> likewise, the REM-HF<sup>14,15</sup> trial using a similar approach was also negative.

Weight may not be a specific enough marker of ADHF, since it may vary for many reasons. It is possible that current markers such as symptoms and weight gain are late and indirect measures of decompensation and that earlier detection of congestion could prompt interventions and avert the incoming ADHF and hospital admission.<sup>15</sup> Monitoring of intrathoracic impedance (Optivol® CRT-D), with an imbedded feature in some of the implanted devices (pacemaker or defibrillator) showed promise, but the DOT-HF study using intrathoracic impedance with an audible alert did not improve outcomes and increased HF admissions,<sup>16</sup> while the recent Multisense trial was negative.<sup>17</sup> Likewise neutral results were observed in stable patients using electronic implanted devices from multiple providers.<sup>14</sup>

Using more sensitive physiologic markers for the development of acute decompensation, such as increased filling pressure, may be beneficial. A variety of implantable hemodynamic monitors (IHM) have been developed to provide objective and continuous information on hemodynamic status in ambulatory HF patients, which may facilitate the timeliness of interventions and improve outcomes. Interesting initial results were obtained for a pacemaker-like device with a RV lead that contains a sensor near its tip to measure right ventricle (RV) pressures (estimated pulmonary artery diastolic (ePAD)) in 274 patients enrolled in the COMPASS HF trial (Chronicle Offers Management to Patients with Advanced Signs and Symptoms of HF). Safety (8% complications, mostly lead dislodgements) and primary efficacy (21% decreased in HF-related events) endpoints were met. Unfortunately, the REDUCE-HF trial (REducing Decompensation events Utilizing intraCardiac prEssures in patients with cHF) was prematurely terminated due to sensor lead failure after 400 patients were enrolled and showed no significant difference in HF events after one year of follow-up. Another device, the Heart-POD (Abbott Laboratories, Illinois, USA) measures directly the left atrial pressure and has shown promising results in a preliminary observational study of 40 ambulatory HF patients. In order to try to further empower the patients in


HOMEOSTASIS, they followed a physician-directed therapeutic strategy guided by left atrial pressure (LAP), which led to a drop in mean daily LAP, decreased the HF hospitalization rate, and resulted in improvements in New York Heart Association (NYHA) class, left ventricular ejection fraction (LVEF) and pharmacological profiles. A larger unblinded study, the LAPTOP-HF trial, 22,23 was recently stopped early due to excess of procedure related complications after enrolment of 486 of the 730 planned patients; the annualized HF hospitalization rates for implanted patients was 0.40 versus 0.68 in Control patients, RRR 41%, p=0.005, offering insights into the benefits of hemodynamic monitoring and the use of physician directed, patient self-management. The patient self-management features have been embedded in a smart phone application that will be available commercially before the end of 2019 and that we propose to use for this protocol.

Recently the FDA and Health Canada approved a novel implantable sensor inserted into the right pulmonary artery that measures pulmonary artery pressures (PAP) in patients with HF, the CardioMEMS<sup>TM</sup> HF System (Abbott Laboratories, Illinois, USA). The coil and capacitor are housed within the sensor to form a miniature electrical circuit that resonates at a specific frequency; variation in PAP will alter the baseline resonant frequency emitted by the sensor, which is electromagnetically coupled to an external antenna for data transmission. Frequency shifts are displayed as pressure waveforms. The data can then be transmitted to the web-based platform for clinical analysis. 24 The CHAMPION trial evaluated the effect of PAP-guided therapy on HFrelated hospitalizations compared to standard of care in 550 patients with NYHA functional class III or IV symptoms. A 28% reduction in HF-related hospitalizations was observed after 6-months of follow-up. 25 As expected, the presence of PH identified HF patients at risk for adverse outcomes, but knowledge of hemodynamic variables allowed for more effective treatment strategies to reduce hospitalizations, albeit with no impact on mortality.<sup>26</sup> Interestingly, both patients with HF with preserved ejection fraction (HFpEF) (using a definition of LVEF > 40%) and HF with reduced ejection fraction (HFrEF) derived benefit,<sup>27</sup> making the CardioMEMS<sup>TM</sup> HF System the first treatment option to show promise for patients with HFpEF, an increasingly recognized cause of group 2 PH.<sup>28</sup> Moreover, patients with chronic obstructive pulmonary disease (COPD) concomitant with HF also derived benefit from hemodynamic monitoring in CHAMPION.<sup>29</sup> An example of the proposed treatment algorithm is available at the


Annex 1.

Further, data from CHAMPION have shown that PH is underestimated by right heart catheterization (RHC) in nearly 50% of patients with HF.<sup>30</sup> RHC provides a "snapshot" of a patient's hemodynamic profile at a single time point, in a hospital-based setting, which may not reflect real life hemodynamics in other settings. These results are consistent with the ESCAPE trial in ADHF patients, which found that pulmonary artery (PA) catheter-guided care was not superior to traditional clinical assessment of volume in preventing subsequent decompensation.<sup>31</sup> However, levels of certain hemodynamic parameters such as pulmonary capillary wedge pressure (PCWP) and mean PA pressure were predictors of later risk for hospitalization. Full characterization of PH status and guidance for medical management may be best accomplished with recurrent assessment of pressures provided by an implanted hemodynamic monitor (IHM). In CHAMPION, patients with no PH on RHC but PH revealed by the IHM had significantly higher HF hospitalization rates than those without this "occult" PH, <sup>30</sup> suggesting that IHM can provide additional information on the patient's overall risk of HF hospitalization. Further, the use of an IHM such as the CardioMEMS<sup>TM</sup> HF System provides an unique opportunity to fine-tune patient management with its dual capacity of providing daily information on congestion (diastolic PAP) and the severity of PH (systolic and mean PAP).

Lastly, there is increasing evidence that filling pressures may influence the arrhythmia burden; a positive relationship has been demonstrated between changes in intra-cardiac pressures and risk for ventricular tachycardia/ventricular fibrillation (VT/VF).<sup>32</sup> There are several potential mechanisms by which an elevated ventricular pressure could influence the development of arrhythmias: stimulation of neurohormonal activation,<sup>33</sup> increase in sympathetic tone,<sup>34</sup> and aberrant intracellular calcium cycling. In addition, acute diastolic stretch shortens action potential duration and refractoriness, whereas chronic dilatation does not,<sup>35</sup> presumably because of activation of stretch-activated channels.<sup>36</sup> There is an opportunity to evaluate the arrhythmia burden in patients with IHM, including atrial fibrillation (AF), VT/VF and implantable cardioverter defibrillator (ICD) events.

The possibility of remote HF monitoring with the CardioMEMS<sup>TM</sup> HF System opens a new avenue for patients with HF, especially the elderly or those living far away from HF clinics. The use of such high-intensity remote monitoring carries the potential for successful detection of parameter


deviations, tailored therapy, more rigorous follow-up and improved outcomes. Moreover, it has

been shown to be cost-effective not only in CHAMPION<sup>36</sup> but also in a real life setting,<sup>4</sup> mostly

because of reduction in hospital readmissions.<sup>37</sup>

At the Montreal Heart Institute (MHI), during the financial year 2018-19 there were 900 hospital

admissions with a primary diagnosis of heart failure in 716 patients. Of those, 34% were readmitted

within the same financial year and 241 patients had  $\geq 1$  readmission (range: 1-9) (see appendix 2).

Targeting these high-risk patients with technology using pulmonary artery pressure monitoring

could possibly expand our ability at the HFC to treat a larger number of patients remotely, decrease

costly hospital readmissions and hence create a virtual heart failure disease management program

(HFDMP).

Accordingly, we propose a paradigm shift towards disease co-management, using patient remote

hemodynamic data, accessed through a smart phone app, and a virtual HF clinic run by a nurse

clinician specialized in HF with the backup of a HF cardiologist.

2. HYPOTHESIS:

2.1 Primary Hypothesis

Due to the dynamic nature of HF and knowledge that filling pressures can rise rapidly over hours

to days, <sup>20</sup> the capacity of patients to get precise PAP measurements as needed will provide critical

information in a timely manner. Using a personalized strategy will allow for appropriate

adjustments of medications based on current PAP values categorized and accessed via a

smartphone app, which will help curtail increases in left-sided filling pressures and thereby avert

hospitalizations for ADHF. Also providing the patient and nurse clinician access to the patients'

hemodynamic data on a continuous basis could empower patients to take more responsibility in

the management of their disease through engagement and self-learning concerning dietary

indiscretion, fluid and salt restriction that may impact PAP measures. Finally, knowledge of their

PAP may provide reassurance in the event of vague symptoms not directly attributable to HF and

decrease the number of emergency department visits. It may also help in making non-HF diagnoses

by eliminating HF as a cause of dyspnea (i.e bronchitis).


3. STUDY OBJECTIVES

To demonstrate that a virtual Heart Failure Clinic (HFC) based on patient self-management using

PAP remote monitoring is superior to usual care of HFC, leads to decreased: hospital admission

for HF, emergency department consultation and/or unplanned intravenous heart failure therapy

and cardiovascular death, compared to a regular HF clinic, has low device-related complications

and is cost-effective, in NYHA class III and II (requiring diuretics) patients.

4. STUDY ENDPOINTS

4.1 Primary Endpoint

The primary endpoint is the time to first occurrence of any component of the composite event as

adjudicated by the Clinical Event Committee (CEC). Components of the event are: acute

decompensated heart failure that requires emergency department consultation and/or unplanned

intravenous heart failure therapy in an outpatient clinic, or hospital admission for heart failure, or

cardiovascular (CV) death during 12 months of follow-up.

4.2 Secondary Endpoints

4.2.1 Time to the first occurrence of the individual components of the composite endpoint

• Acute decompensated heart failure that requires emergency department consultation

and/or unplanned intravenous heart failure therapy in an outpatient clinic;

Hospital admission for heart failure;

CV death

4.2.2 Changes in functional capacity between baseline and 12-months

NYHA functional class;

Quality of life (Kansas city cardiomyopathy (KCCQ) questionnaire);

• 6 minute walk distance.

4.2.3 Device-related endpoints (for CardioMEMS group only)

Safety: adverse events related to the device;

Number of successful patient contacts (virtual and clinic);

■ PA pressures: changes, frequency of elevated readings;

■ Ease of application utilization.


4.2.4 Cost-effectiveness

A cost utility analysis will be undertaken as part of the study protocol to evaluate the impact

of the treatment strategy of remote PAP monitoring compared to usual care. An incremental

cost-effectiveness ratio (ICER) will be calculated by comparison of calculated costs and

quality-adjusted life years in both study groups. This data will then be used to construct an

economic model to evaluate the cost-effectiveness in a hypothetical cohort of 10,000

patients. This data will be used to calculate the incremental cost per Quality-Adjusted Life

Year (QALY) gained and per life-year gained. We will perform deterministic sensitivity

analyses to explore the impact of uncertainty in key parameters on the analysis results and a

probabilistic sensitivity analysis to further characterize uncertainty in model parameters.

Detailed resource utilization and costs will be collected prospectively for randomized

patients, including diagnostic evaluation costs directly incurred as a result of the

CardioMEMS™ HF System procedure, procedural costs, and inpatient treatment costs at a

large tertiary care hospital in Montreal (MHI). Individual patient-level costs of heart failure

hospitalizations, emergency room (ER) visits, and short stay costs for intravenous diuretics

will be obtained from the Montreal Heart Institute. Follow-up costs will include protocol

driven visits and tests, and additional unscheduled outpatient treatment visits for heart failure

or visits to the HFC.

Evaluation of quality of life will be performed using the KCCQ questionnaire and quality

adjusted life years (life expectancy adjusted for quality of life of the health state experienced)

will be calculated for each patient in the alive state using published health utilities, which

measure quality of life from a 0 (dead) to 1 (perfect health) scale, for heart failure according

to NYHA Class and results of the KCCQ questionnaire. In the absence of questionnaire data

for hospitalized patients, utility decrements will be applied for heart failure hospitalizations

and emergency room visits as per the published literature. A short-term utility decrements

(i.e. disutility) for the CardioMEMS<sup>TM</sup> procedure will be approximated using published

decrements for percutaneous coronary intervention (PCI).


#### 4.3 Tertiary/Exploratory Endpoints

#### 4.3.1 Goal for best practice

- % achieved target dose of Guidelines-derived medical therapy (GDMT) (HFrEF);
- Medication changes (mean dose achieved by class of GDMT) between baseline and 12 months;
- Time (days) to achieve target doses of GDMT (HFrEF).

#### 4.3.2 Changes in echocardiographic parameters between baseline and 12 months

Cardiac remodeling including left ventricle (LV) end-systolic and end-diastolic volumes indexed to blood surface area (BSA), LVEF, RV dimensions and function including RV-PA coupling, left atrium (LA) volume, mitral and tricuspid regurgitation severity, with a complete echocardiography protocol proposal and Core Laboratory analysis.

#### 4.3.3 Changes in biomarkers levels between baseline and 12-months

■ Blood samples will be collected for biomarkers analysis: General (Electrolytes, BUN, creatinine and CBC), and disease-specific (HS-CRP, NT-proBNP, troponin, Osteopontin, Angiotensin-II, aldosterone, ST2, Vasopressin, galectin-3, PIIINP, cystatin C).

#### 4.3.4 Arrhythmia Burden

- Episodes of atrial fibrillation requiring medical attention (ED visits or hospitalization);
- VT/VF events:
- Anti-tachycardia pacing or appropriate ICD shocks in patients with an ICD

#### 4.3.5 Patient quality of life and satisfaction

 Regarding both the virtual follow-up itself and the personalized algorithm using the application. Standardized quality of life questionnaires will be used.

#### 4.3.6 Drug concentrations

■ Blood samples will be collected to measure concentrations of drugs commonly used in HF patients at the baseline visit, as well as at visits at week 2, month 2, month 12 and at unscheduled visits.


5. STUDY PROTOCOL

5.1 Study design

Type of study: A single center prospective randomized open-label blinded-endpoint (PROBE) trial

is proposed comparing two strategies for patients with HF who had at least one admission for a

primary diagnosis of HF regardless of LVEF in the previous year i.e., usual care by a specialized

multidisciplinary HF clinic team versus hemodynamic monitoring and self-empowered remote

follow-up using the newly developed smart-phone/iPad application, with the back-up of a nurse

clinician and a HF cardiologist and limited HF clinic visits.

150 eligible patients who consent to participate will be randomized to the control group or

intervention group in a 1:1 ratio. Patients randomized to hemodynamic monitoring (CardioMEMS

group) will have the CardioMEMS<sup>TM</sup> HF System implanted as an outpatient procedure within a

week of random assignment.

Before randomization, patients will need to be stable as judged by the treating HF clinic

cardiologist. After randomization, all subjects will receive education on HF as per local practice

as well as recommendations regarding nutrition and exercise, for daily weights, medication

record, clinical notes and appointments.

Patients in the control group will be followed as per usual practice by the MHI multidisciplinary

HF clinic. Patients in the CardioMEMS group will be seen at baseline, week 1 and week 2 after

implantation, two months and twelve months after randomization and will be in regular contact

with the lead research nurse with virtual follow-ups at weeks 3, 4, 6, 12, 16, 20, 24, 28, 32, 36, 40,

44, and 48. The specialized HF clinician nurse and cardiologist will design an individualized pre-

specified therapeutic plan according to CHF guidelines and clinical experience with that individual

patient (Appendix 3). For HFrEF, GDMT will be implemented in both groups, including ICD and

CRT referral when indicated.

For patients in the CardioMEMS group, a blood pressure cuff will be provided and hemodynamic

data will be taken twice daily by the patient from the moment of randomization in the trial. i-Pad®

internet communication using Skype/Facetime or telephone calls will be done twice in the first

month, once in the second month and monthly thereafter, unless a medical problem occurs that


requires more frequent contact, which will be determined by the study team. The patient will implement the individualized therapeutic plan designed by the HF clinician nurse and cardiologist, following a pre-specified algorithm (Appendix 1), which includes titration of angiotensinconverting enzyme (ACE) inhibitors, angiotensin receptor blockers (ARB), angiotensin receptor neprilysin inhibitors (ARNI), hydralazine, nitrates, beta-blockers and mineralocorticoid antagonists as needed. Initiation of some of these medications may require a visit to the research clinic, if judged necessary and will be counted as unscheduled visit. Diuretics and potassium supplementation will be adjusted according to individualized target PAP pressures, electrolytes and renal function. Blood samples for electrolytes and renal function: sodium, potassium, chloride, and bicarbonate will be drawn one week after any changes of medications, or as deemed clinically indicated by the treating team. The research team will follow the laboratory results and intervene as needed. Objectives for PAP pressures will be similar to the CHAMPION trial, i.e., PAP systolic (15–35 mmHg), PAP diastolic (8–20 mmHg), and PAP mean (10–25 mmHg). PA measurements will be transmitted daily for the first two weeks, three times a week thereafter, and more frequently as needed. Also, patients will have access to the research nurse coordinator for advices or to signal changes in their state (for example a bronchial infection, diarrhea etc.). Further, patients in the CardioMEMS<sup>TM</sup> group will have access to categorized data (very low, low, in range, high or very high pressures) using the app and be able to adjust their medication (mostly diuretics) according to an individualized algorithm. Furthermore, data reaching thresholds will be reviewed daily during working days and patients will be contacted in the event of clinically significant changes, as individually defined at the outset. The general aim is to introduce and rapidly up-titrate GDMT for patients with HFrEF (ACEi, ARB or ARNI), beta-blockers and mineralocorticoid receptor antagonists (MRA), to reduce or eliminate diuretic doses for patients with low or very low PAP, and to increase diuretic or vasodilator doses for high or very high PAP. A general algorithm is proposed in Appendix 1.

#### 5.2 Inclusion/Exclusion Criteria

#### 5.2.1 Inclusion Criteria

- 1. Male or female  $\geq$  18 years old.
- Symptomatic HF (NYHA III) with recent heart failure admission in the previous year (12 months). OR


3. Patient with at least one ER visit or unplanned HF clinic requiring iv diuretics within 12 months will be eligible if they have in addition a N-terminal pro-BNP (NT-proBNP) level > 800pg/ml at screening <u>AND</u> NYHA Class II on diuretics (furosemide ≥ 40mg qd), III or ambulatory IV.

4. HF with reduced or preserved EF of at least 3 months duration.

5. Minimum technological knowledge either with a smartphone or iPAD for use of the self-management application, including access to internet.

6. Anatomical criteria

a. PA branch diameter between 7 mm – 15 mm

b. For BMI >35, distance from patient's back to target PA<10cm

**5.2.2** Exclusion Criteria

In order to maximize the generalizability of the results, exclusion criteria will be kept to a minimum:

1. *Recent cardiovascular event*: Acute coronary syndrome (STEMI/NSTEMI; a small rise in the troponin level would be expected in this population and is not a contraindication for enrolment); Percutaneous Coronary Intervention (PCI), new cardiac rhythm management (CRM) device (pacemaker, ICD and CRT), CRM system revision, lead extraction or cardiac or other major surgery or transient ischemic attack or stroke within 2 months (3 months of stabilization after CRT or cardiac surgery);

2. Scheduled cardiac surgery;

3. History of pulmonary embolism or recurrent deep vein thrombosis;

4. Persistent NYHA Class IV and ACC/AHA HF Stage D, patients implanted with a ventricular assist device (VAD), or patients listed for cardiac transplantation and likely to be transplanted within 12 months;

5. Coexisting severe stenotic valve lesions, endocarditis, obstructive hypertrophic cardiomyopathy, acute myocarditis, tamponade, or large pericardial effusion;

6. Clinically too unstable to be followed remotely; this includes but is not limited to:

a. Resting systolic blood pressure < 80 or > 180 mmHg;

b. Resting heart rate > 100 bpm;

- c. Stage IV or V chronic kidney disease (Estimated Glomerular Filtration Rate (eGFR) that remains < 30 mL/min/1.73m<sup>2</sup> by MDRD) or nonresponsive to diuretic therapy or on chronic renal dialysis;
- 7. Severe pulmonary hypertension with systolic pulmonary artery pressure ≥80 mmHg;
- 8. Pulmonary hypertension other than group II PH;
- 9. Anemia requiring transfusions, iron infusions, or hemoglobin below 100;
- 10. Coagulopathy or uninterruptible anticoagulation therapy or contraindication to antiplatelet/anticoagulant treatments anticipated in the protocol;
- 11. Intolerance to aspirin or clopidogrel;
- 12. Active infection requiring systemic antibiotics;
- 13. Unwillingness to sign informed consent or to attend the outpatient clinic;
- 14. Participation in another research trial with intervention;
- 15. Discharge to a chronic care facility or residence in an outlying area;
- 16. Pregnant or lactating women or women of childbearing potential who are not protected from pregnancy by an accepted method of contraception, such as the oral contraceptive pill, an intrauterine device or surgical sterilization. If necessary a negative urine or blood test will be performed before randomization
- 17. Any condition that in the opinion of the investigator would jeopardize the evaluation for efficacy or safety or be associated with poor adherence to the protocol, including cognitive decline.
- 18. Life expectancy <1 year;

#### 5.3 Subject Attribution Number

Once informed consent is obtained, each subject will be assigned a unique 3-digit subject identification (SID) number ("Subject number") for unambiguous identification throughout the study; it will be constructed as follows:

3 Digits: Subject number, unique within the study center starting at 001.

Sequential numbers will reflect the order in which subjects are recruited. SID numbers will be used in sequence with no number skipped, substituted, or re-used.


6. SUBJECT EVALUATION

**6.1 Informed Consent** 

Before any screening examination takes place, potentially eligible subjects will be given a full

explanation as to what the study entails. This will be performed verbally and in writing. Subjects

will be given ample time to consider participation and pose any questions they may have. Subjects

who are willing to take part in the study will then be asked to sign an informed consent form.

Screening examinations will only be performed after written informed consent is obtained.

Subjects who continue to meet enrolment criteria upon completion of the screening process will

be eligible for randomization.

6.2 Visits

At Baseline visit the consent form will be signed and inclusion and exclusion criteria will be

reviewed before randomization. Only Baseline and Final Visits will be scheduled in the study for

the Control Group. All other visits will be scheduled according to usual care by the treating HF

clinic team.

**Baseline visit** (Visit 1)

Informed Consent

Allocation of unique SID number

Demographic information: demographic data and other population characteristics including

sex, race, year of birth, age, smoking history, and alcohol consumption

Medical and surgical cardiovascular history (including cardiovascular risk factors)

NYHA Class

Physical examination by physician

• Vital signs in sitting position (blood pressure (BP) and heart rate (HR)) after resting for at

least 5 min, 2 measurements, 2 minutes apart

Weight, height

Echocardiography

• 12-lead ECG in supine position, after resting for at least 5 min.

Assessment of eligibility criteria

Randomization to study group


- Current therapy and timing
- Subject education: nutrition, exercise, education regarding HF
- Blood tests
  - o BUN, Creatinine, Electrolytes, CBC, NT-proBNP
  - Blood samples for subsequent analysis: Cystatin-C, Angiotensin-II, Aldosterone,
     Vasopressin, hS-CRP, ST2, Galectin-3, Troponin, Osteopontin, PIIINP, drug
     concentrations.
- Urine or blood pregnancy test for women of childbearing potential
- 6-minute walk test
- Quality of Life Questionnaire (MLHF)

#### For patients randomized to CardioMEMS:

#### **Implantation Visit** (visit 2)

- CardioMEMS Implantation
- Hemodynamic data collection
- Assessment of AEs/SAEs

#### Week 1 after implantation (Visit 3)

- Adjustment of medication
- Subject technology training
- Assessment of AEs/SAEs

#### Week 2 after implantation (Visit 4)

- NYHA Class
- Physical examination by physician
- Vital signs in sitting position (blood pressure (BP) and heart rate (HR)) after resting for at least 5 min, 2 measurements, 2 min apart
- Weight
- Current therapy and timing
- Adjustment of medication
- Lab Assessment : BUN, Creatinine, Electrolytes, CBC, NT-ProBNP


- Blood sample for drug concentrations
- Assessment of AEs/SAEs

#### Month 2 (Visit 5)

- NYHA Class
- Physical examination by physician
- Vital signs in sitting position (blood pressure (BP) and heart rate (HR)) after resting for at least 5 min, 2 measurements, 2 min apart
- Weight
- Current therapy and timing
- Adjustment of medication
- Lab Assessment: BUN, Creatinine, Electrolytes, CBC, NT-proBNP
- Blood sample for drug concentrations
- Assessment of AEs/SAEs

#### **Virtual Visits**

Virtual visits will be done remotely (patient self-management using PAP monitoring) following hospital discharge of the implant: week, 3, 4, 6, 12, 16, 20, 24, 28, ..., 48

- Current therapy
- Adjustment of medication
- Remote evaluation by nurse: HF symptoms
- Remote hemodynamic evaluation by nurse
- Laboratory assessment (if clinically indicated 1 week after change in medication dosage)
- Assessment of AEs/SAEs

#### For all randomized patients:

#### **Unscheduled Visit(s)**

- NYHA Class
- Physical examination by physician
- Vital signs in sitting position (blood pressure (BP) and heart rate (HR)) after resting for at least 5 min, 2 measurements, 2 min apart


- Weight
- 12-lead ECG (if indicated).
- Current therapy and timing
- Adjustment of medication
- Blood tests
  - o BUN, Creatinine, Electrolytes, CBC, NT-proBNP
- Blood samples for drug concentrations
- Assessment of AEs/SAEs

#### Month 12 (Final Visit 6)

- NYHA Class
- Changes in medical and surgical cardiovascular history
- Physical examination by physician
- Vital signs in sitting position (blood pressure (BP) and heart rate (HR)) after resting for at least 5 min, 2 measurements, 2 min apart
- Weight
- Echocardiography
- 12-lead ECG in supine position, after resting for at least 5 min.
- Current therapy and timing
- Blood tests: BUN, Creatinine, Electrolytes, CBC, NT-proBNP
- Blood samples for subsequent Analysis: Cystatin-C, Angiotensin-II, Aldosterone,
   Vasopressin, hs-CRP, ST2, Galectin-3, Troponin, Osteopontin, PIIINP, drug concentrations.
- 6 minute walk test
- Quality of Life Questionnaire (MLHF)
- Assessment of AEs/SAEs

#### **End of study visit:**

Every implanted participant will be followed at the Heart Failure Clinic at the end of the trail within one month of study termination.


#### 7. FLOW CHART

| | CardioMEMS and CONTROL GROUPS | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Group | Both Groups | CardioMEMS Group Only | | | | | | Both Groups |
| Visit (V) | Baseline Randomization Visit 1 | Implantation<br>Visit 2 | Week 1 post implantation Visit 3 | Week 2 post implantation Visit 4 | Month 2 (5)<br>Visit 5 | Virtual <sup>(5)</sup><br>Week 3, 4, 6,12, 16<br>20,24,28,,48 | Unscheduled | Month 12 (5) Final visit Visit 6 |
| Visit Windows (days) | 0 | ≤7 | ±4 | ±4 | ±14 | ±4 | | ±14 |
| Informed Consent Form | X | | | | | | | |
| Demographics | X | | | | | | | |
| Medical & Surgical CV History | X | | | | | | | $X^6$ |
| NYHA Class | X | | | X | X | | X | X |
| Physical Exam by physician | X | | | X | X | | X | X |
| Vital Signs | X | | | X | X | | X | X |
| Weight | X | | | X | X | | X | X |
| Height | X | | | | | | | |
| Echocardiography | X | | | | | | | X |
| ECG | X | | | | | | X (3) | X |
| Inclusion/Exclusion criteria | X | | | | | | | |
| Randomization to Study Group | X | | | | | | | |
| Current Therapy and timing | X | | | X | X | X | X | X |
| Adjustment of Medication | | | X | X | X | X | X | X |
| Subject Education (Nutrition, exercice etc.) | X | | | | | | | |
| CardioMEMS Device | | X | | | | | | |
| Subject Technology Training | | | X | | | | | |
| Remote evaluation by nurse: HF symptoms | | | | | | X | | |
| Remote hemodynamic Evaluation by nurse: | | | | | | X | | |
| Hemodynamic Data Collection | | X | | | | | | |
| Laboratory Assessment: Electrolytes,<br>Creatinine, CBC, Urea, NT-proBNP | X | | | X | X | | X | X |
| Laboratory Assessment (Virtual Visit): | | | | | | X (4) | | |
| Blood sample for subsequent analysis: Cystatin C, Angiotensin-II, Aldosterone, Vasopressin, HS-CRP, Galectin-3, Troponin. Osteopontin, ST2, PIIINP | X | | | | | | | X |
| Urine Pregnancy Test | $X^{(1)}$ | | | | | | | |
| Drug concentrations | X | | | X | X | | X | X |
| 6 min walk test | X | | | | | | | X |
| Quality of Life Questionnaire (KCCQ) <sup>2</sup> | X | | | | | | | X |
| Assessment of AEs/SAEs | | X | X | X | X | X | X | X |

<sup>(1)</sup> For women of childbearing potential (2) Kansas City Cardiomyopathy Questionnaire


<sup>(3)</sup> If indicated (5) Post baseline visit (6) Change(s) in Med & Surgical CV History (4) No Blood test except by local lab if clinically indicated (1 week after change in medication dosage)

7. SPECIFIC ASSESSMENTS

7.1 End point variables

Blood pressure measurement, biochemistry monitoring and renal function

Blood pressure will be measured and recorded at each visits according to the recommendations of

the Canadian Hypertension Education Program.<sup>38</sup> Electrolytes, serum creatinine and vital signs

will be assessed as described in the Study flow chart. In the assessment renal function, eGFR will

be calculated as previously described using the MDRD equation.<sup>39</sup>

Cystatin C

Moreover, in order to better characterize changes in renal function during the study, cystatin C will

be measured at baseline and at the end of the study. Cystatin C is a novel biomarker of renal

function which appears to be more sensitive than serum creatinine to detect modest changes in

renal function. <sup>40</sup>Moreover, in HF, it has been shown to be a powerful prognostic marker. <sup>40</sup>

N-terminal proB-type natriuretic peptide (NT-proBNP).

BNP is secreted primarily from the ventricles in both healthy individuals and patients with CHF.<sup>41</sup>

The production of BNP in the ventricle increases proportionally with increases in both ventricular

wall tension and stretch. Both BNP and NT pro-BNP, the inactive portion of pro-BNP, have been

shown to correlate with LVEF, left ventricular volumes and pressures. While neurohumoral

blockade decrease the NT-proBNP levels and prognosis, to our knowledge, there has been no study

showing that effective pressure management significantly reduce concentrations of BNP and NT-

proBNP. NT-proBNP will be measured by Dr. Joel Lavoie using the « Roche proBNP assay »

(Roche Diagnostics, Mannheim, Germany), on the Elecsys 2010 analyzer (Roche diagnostics).

Our group has had extensive experience in measuring NT-proBNP in previous studies. 42-45

PHINP

It is now widely accepted that aldosterone induces deleterious effects on extracellular matrix

balance, for which type I and III collagen constitute the majority of the collagen. 46-48 These

alterations in collagens type I and III have been proposed to play a key role in myocardial

stiffness. 48 Previous work has demonstrated that PIIINP serum levels were associated with poor

outcomes in patients with HF. 49,50 Because it is expected that pressure management will reduce


myocardial stress in HF patients,50-52 PIIINP will also be measured. PIIINP will be measured in

the laboratory at the Montreal Heart Institute directed by Dr Martin G. Sirois using the Orion

Diagnostica's UniQ PIIINP assay. The use of this assay has been validated in numerous studies in

humans. Dr Sirois's laboratory has measured PIIINP in a study comparing circulating levels of

various biomarkers between patients with systolic HF and HF-PEF, as well as in a study comparing

concentrations of biomarkers between patients with HF and anemia and HF patients without

anemia.<sup>53</sup> Together with NT-proBNP, this biomarker will be very important in demonstrating that

the beneficial effects of pressure management on cardiac remodeling.

Osteopontin (OPN)

An additional marker of remodeling, osteopontin [OPN]) is a glycoprotein that can be detected in

plasma and was found to be upregulated in several animal models of cardiac failure<sup>54</sup> and may thus

represent a new biomarker that facilitates risk stratification in patients with heart failure;<sup>48</sup> it has

been shown to correlate with disease severity and poor prognosis. 55,56 OPN seems to have a pivotal

role in the development of Angiotensin II-induced cardiac fibrosis and remodeling. Moreover, the

effect of Eplerenone on the prevention of cardiac fibrosis, but not cardiac hypertrophy, might be

partially mediated through the inhibition of OPN expression.<sup>57</sup> Thus, we will also measure

angiotensin-II and aldosterone, two important steps in the remodeling and fibrosis pathways.

**High sensitivity C-Reactive protein (HS-CRP)** 

While heart failure has been shown to be an inflammatory condition, <sup>58,59</sup> the impact of pressure

management on HS-CRP has not been well characterized. We herein propose to measure HS-CRP

in our patients undergoing hemodynamic monitoring.

Cardiac Troponin T (cTnT)

In heart failure, the level of troponin correlates with prognostic independently of the presence of

ischemic etiology or myocardial stretch assessed by NT-proBNP. This troponin leak varies with

time and has been shown to be associated with decreased survival. We herein propose to measure

cTnT in our patients undergoing hemodynamic monitoring.


**Emerging markers** 

Galectin-3 serves important functions in numerous biological activities including cell growth,

apoptosis, pre-mRNA splicing, differentiation, transformation, angiogenesis, inflammation,

fibrosis and host defense. 60-63 Numerous previous studies have indicated that galectin-3 may be

used as a diagnostic or prognostic biomarker for certain types of heart disease, kidney disease and

cancer. <sup>64</sup> Galectin-3 levels are correlated with elevated risk for new HF in healthy people and acute

myocardial infarction with reduced ejection fraction patients.<sup>65</sup> Thus, it is probable that galectin-

3 has a more important role in the beginning stage of HF including early fibrosis and ventricular. <sup>66</sup>

Whether hemodynamic management leads to improved levels of the biomarker is unknown at the

present time.

ST2 cardiac biomarker is a protein biomarker of cardiac stress encoded by the IL1RL1 gene.

ST2 signals the presence and severity of adverse cardiac remodeling and tissue fibrosis, which

occurs in response to myocardial infarction, acute coronary syndrome, or worsening heart

failure. 62,67,68,59 ST2 provides prognostic information that is independent of other cardiac

biomarkers such as BNP, NT-proBNP, highly sensitive troponin, GDF-15, and galectin-3.<sup>[3]</sup> One

study indicated that discrimination is independent of age, body mass index, history of heart

failure, anemia and impaired renal failure or sex.

Vasopressin (arginine vasopressin, AVP; antidiuretic hormone, ADH) is a peptide hormone

formed in the hypothalamus, then transported via axons to the posterior pituitary, which releases

it into the blood. AVP has two principle sites of action: the kidney and blood vessels. <sup>69</sup> The primary

function of AVP in the body is to regulate extracellular fluid volume by regulating renal handling

of water, although it is also a vasoconstrictor. AVP acts on renal collecting ducts via V<sub>2</sub> receptors

to increase water permeability (cAMP-dependent mechanism), which leads to decreased urine

formation (hence, the antidiuretic action of "antidiuretic hormone"). This increases blood volume,

cardiac output and arterial pressure. Heart failure is associated with what might be viewed as a

paradoxical increase in AVP. Increased blood volume and atrial pressure associated with heart

failure should decrease AVP secretion, but it does not. It may be that sympathetic and renin-

angiotensin system activation in heart failure override the volume and low pressure cardiovascular


receptors (as well as the hypothalamic control of AVP release) and cause an increase in AVP

secretion. 70 Nevertheless, this increase in AVP during heart failure may contribute to the increase

in systemic vascular resistance as well as the enhanced renal retention of fluid that accompanies

heart failure. Whether hemodynamic monitoring leads to a decrease in AVP is unknown.

**Drug concentrations** 

Concentrations of commonly used drugs in patients with HF will be measured at the baseline visit,

as well as at visits at week 2, month 12 and at unscheduled visits. At each of these visits,

the dose, the time of administration of the last dose of the cardiovascular medications and the time

of the blood draw will be recorded.

Currently, very little information is available regarding the pharmacokinetic (PK) or

concentrations of drugs in HF patients.<sup>71</sup> Data from our group and others have suggested marked

differences in the concentrations or PK of commonly used drugs in HF patients compared to

healthy individuals such as spironolactone and candesartan (manuscripts submitted). This could

be attributable to several factors such as decreased renal function. 71 Moreover, only very limited

data are available on the factors influencing the PK of drugs in patients with HF.<sup>71</sup>

In addition, little information is available on the magnitude of the effects of common dosing

adjustments of HF drugs in "real-life" HF patients on drug concentrations, or whether patients who

cannot reach target doses of HF medication actually have lower drug concentrations than those

who do. Indeed, some patients who do not reach target doses could present comparable drug

concentrations as patients reaching target doses, if they present clinical factors that predispose to

increased concentrations, such as renal dysfunction.<sup>71</sup>

The screening and quantification of drugs or their active metabolites will be performed in plasma

at the Platform of Biopharmacy of the Faculty of Pharmacy at Université de Montréal using Liquid

Chromatography coupled to triple quadrupole mass spectrometer (LC-MS/MS) in the selective

MRM mode<sup>72-76</sup> and Liquid Chromatography High-Resolution Mass Spectrometer (LC-HRMS)

of the type quadrupole time-of-flight (QTof) in the full scan mode. <sup>77-82</sup> This group has an extensive

experience for developing and optimising the bioanalytical techniques needed to measure

drugs/metabolites.83-97 In addition to comparing drug concentrations between groups and

concentrations changes, for drugs used in 30 or more patients, we will perform exploratory

population-pharmacokinetics modelling. Modelling analyses will be performed by the STP2

Laboratory (Faculty of Pharmacy at Université de Montréal) using the gold standard for population

pharmacokinetics modelling to estimate parameter and, interindividual and residual variability. 98,99

Population pharmacokinetics modelling will be done using nonlinear mixed effect modeling

(NONMEM®, version 7.4, ICON Development Solutions). Pharmacokinetics studies in patients

with special conditions are at the center of the STP2 Laboratory research. 100-108

8. SAFETY

All Adverse events and serious adverse events will be reviewed by the investigator or a sub-

investigator.

8.1. Definition of Adverse Events, Serious Adverse Events, and procedures for reporting

**Serious Adverse Event** 

8.1.1. Adverse Event (AE)

An AE is any untoward medical occurrence, unintended disease or injury, or untoward

clinical signs (including abnormal laboratory findings) in subjects, users or other persons,

whether or not related to the investigational medical device.

This definition includes events related to the investigational medical device and events

related to the procedures involved.

8.1.2. Serious Adverse Event definition (SAE)

A serious adverse event is an AE that fulfills one or more of the following:

1. Results in death

2. Led to serious deterioration in heath of the subject, that either resulted in

• A life-threatening illness or injury, or

• A permanent impairment of a body structure or a body function, or

• Requires in-patient hospitalization or prolongation of existing hospitalization


Medical or surgical intervention to prevent life-threatening illness or injury or

permanent impairment to a body structure or a body function

3. Results to fetal distress, fetal death or a congenital abnormality/birth defect.

Note: Planned hospitalization for a pre-existing condition or a procedure is not considered

a serious adverse event.

8.1.3. Adverse device Effect (ADE)

Adverse event related to the use of an investigational medical device.

Notes: This definition includes adverse events resulting from insufficient or inadequate

instructions for use, deployment, implantation, installation, or operation, or any

malfunction of the investigational medical device.

This definition includes any event resulting from use error or from intentional misuse of

the investigational medical device.

8.1.4. Serious Adverse Device Effect (SADE)

Adverse device effect that has resulted in any of the consequences characteristic of a

serious adverse event

8.1.5. Unanticipated Serious Adverse Device Effect (USADE)

Any serious adverse effect on health or safety or any life-threatening problem or death

caused by, or associated with, a device, if that effect, problem, or death was not previously

identified in nature, severity, or degree of incidence in the CardioMEMS user's Manual, or

any other unanticipated serious problem associated with a device that relates to the rights,

safety, or welfare of subjects <sup>41</sup>

8.1.6. Procedures for Adverse Event reporting

8.1.6.1. Investigator Reporting

All AEs considered device related will be recorded in the eCRF for enrolled subjects.


Any Serious Adverse Event that occurs in the course of the study must be reported to

Montreal Health Innovations Coordinating Center (MHICC) within one day of the

investigator becoming aware of the SAE. All SAEs will be recorded in the electronic Case

Report Form (eCRF) as adverse events up to 14 days after final visit. The investigator is

responsible for informing the Ethics Committee of the SAE as per local requirements.

9. STATISTICAL ANALYSIS

Descriptive statistics of all study endpoints will be presented overall and broken down by group.

Number of observations, mean, standard deviation, median, minimum and maximum will be

presented for continuous variables. Count and proportion will be displayed for categorical

variables.

For the primary endpoint, the analysis will consist of an unadjusted comparison of time to first

event. Event-rate curves will be estimated by the Kaplan-Meier product-limit method and the

difference between groups will be assessed using the log-rank test. Components of the primary

endpoint will be analyzed similarly.

ANCOVA models will be used to compare continuous endpoints expressed as change from

baseline to 12 months between the standard group and the virtual group. The main model will

include fixed effects for group with the baseline value as a covariate. Difference between groups

in other continuous endpoints will be tested by either two-sample t-tests or Wilcoxon rank-sum

tests depending on the normality of the data. Difference between groups in categorical endpoints

will be tested using Chi-square tests.

Basic assumptions of the proposed analyses will be checked and data transformation or other

analyses could be done if appropriate. For example, as some endpoints are likely to be skewed (ex.

hs-CRP), log-transformation might be used, in which case descriptive statistics would also include

geometric means. Missing values will not be imputed.

All statistical tests will be two-sided and conducted at the 0.05 significance level. Statistical

analyses will be done using SAS version 9.4 or higher.


A statistical analysis plan (SAP) will be written to fully describe the statistical analyses that will

be done. The SAP will be finalized prior to database lock.

9.1. Sample size

It is hypothesized that virtual monitoring will be superior to standard care in reducing the risk of

the composite primary endpoint of acute decompensated heart failure that requires emergency

department consultation and/or unplanned intravenous heart failure therapy in an outpatient clinic,

hospital admission for heart failure, or CV death during 12 months of follow-up. The sample size

rationale and assumptions are based on the following:

From the CHAMPION trial, the rate of HF hospitalization at 12 months was 0.52 and 0.75 in the

treatment and control groups respectively (Phil Adamson personal communication, unpublished

data), leading to a hazard ratio of 0.53. Similar event rates are expected for the primary endpoint

in this trial. The mortality rate is expected to be similar between the two groups as in CHAMPION.

Using a log-rank test, a total of 136 subjects (68 in each group) would provide 80% power with a

two-sided significance level of  $\alpha$ =0.05. Factoring in a drop-out rate of approximately 10%, a total

of 150 patients are required.

10. INVESTIGATOR'S REGULATORY OBLIGATIONS

10.1. Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approval

The protocol and the informed consent document must have the initial and at least annual (when

required) approval of an IRB/IEC. The signed IRB/IEC approval letter must identify the

documents approved (i.e. list the investigator's name, the protocol number and title, the date of the

protocol and informed consent document, and the date of approval of the protocol and the informed

consent document). Written information to be provided to the subject (i.e. patient cards, patient

diary, instructional material on nutrition, exercise, and HF) and any advertisement used to recruit


subjects must also be reviewed by the IRB/IEC.

10.2. Informed Consent

Regulatory agencies have issued regulations to provide protection for human subjects in clinical

investigations and to describe the general requirements for informed consent. The informed

consent document shall contain all the elements of informed consent specified in the application

regulations. Some regulations may require the disclosure of additional information to the subject

and/or inclusion of additional information in an informed consent document.

10.3. Declaration of Helsinki

This study will be conducted in accordance with the ethical principles that have their origin in the

Declaration of Helsinki (Appendix 5) and that are consistent with good clinical practices (GCP)

and the applicable requirements.

10.4. Case Report Form

All data will be recorded on eCRF provided by the MHICC.

10.5. Confidentiality

All records identifying the subject will be kept confidential and, to the extent permitted by the

applicable laws and/or regulations, will not be made publicly available.

Subject names will not be supplied. Only the subject number will be recorded in the eCRF, and if

the subject name appears on any other document (e.g. pathologist report), it must be obliterated

before a copy of the document is supplied to the sponsor. Study findings stored on a computer will

be stored in accordance with local data protection laws. As part of the informed consent process,

the subjects will be informed in writing that representatives of the sponsor, IEC/IRB, or regulatory

authorities may inspect their medical records to verify the information collected, and that all

personal information made available for inspection will be handled in strictest confidence and in

accordance with local data protection laws.

If the results of the study are published, the subject's identity will remain confidential.

The investigator will maintain a list to enable subjects to be identified.


11. DATA QUALITY ASSURANCE

The principal investigator performs quality control and assurance checks on all clinical studies that

he/she performs. Before enrolling any subjects in this study, the principal investigator and study

coordinator review the protocol and the eCRFs, determine the procedure for obtaining informed

consent, and determine the procedure for reporting AEs and SAEs. The principal investigator or

study coordinator reviews the data for accuracy and safety information. The principal investigator

or study coordinator reviews the data for legibility, completeness and logical consistency.

11.1. Monitoring, Audits and inspections

In accordance with applicable regulations, GCP, and sponsor's / Academic Contract Research

Organization's (ARO) procedures, monitors will contact the site prior to the start of the study to

review with the site staff the protocol, study requirements, and their responsibilities to satisfy

regulatory, ethical, and sponsor's requirements. When reviewing data collection procedures, the

discussion will also include identification and documentation of source data items.

The sponsor's designee will monitor the site activity to verify that the:

Data are authentic, accurate, and complete

Safety and rights of subjects are being protected

Study is conducted in accordance with the currently approved protocol (including study

procedures in accordance with the protocol)

Any other study agreements, GCP, and all applicable regulatory requirements are met.

The investigator and the head of the medical institution (where applicable) agrees to allow the

monitor direct access to all relevant documents.

To ensure compliance with GCP and regulatory requirements, a member of the sponsor's (or a

designated ARO's) quality assurance unit may arrange to conduct an audit to assess the

performance of the study at the study site and of the study documents originating there. The

investigator / institution will be informed of the audit outcome.

In addition, inspections by regulatory health authority representatives and IEC(s) / IRB(s) are

possible. The investigator should notify the MHICC immediately of any such inspection.


The investigator / institution agrees to allow the auditor or inspector direct access to all relevant

documents and allocate his / her time and the time of his / her staff to the auditor / inspector to

discuss findings and any issues. Audits and inspections may occur at any time during or after

completion of the study.

11.2. Archiving

Essential documents shall be archived safely and securely in such a way that ensures that they are

readily available upon authorities' request.

Patient (hospital) files will be archived according to local regulations and in accordance with the

maximum period of time permitted by the hospital, institution or private practice. Where the

archiving procedures do not meet the minimum timelines required by the sponsor, alternative

arrangements must be made to ensure the availability of the source documents for the required

period.

The investigator/institution notifies the sponsor if the archival arrangements change (e.g.

relocation or transfer of ownership).

The investigator site file is not to be destroyed without the sponsor's approval.

The investigator's contract will contain all regulations relevant for the study center.

12. DATA MANAGEMENT

The MHICC will be the data coordinating center. The data collection tool for this study will be a

validated electronic system. Subject data necessary for analysis and reporting will be entered into

database or data system. Clinical data management will be performed in accordance with

applicable sponsor's standards and data cleaning procedures. This is applicable for data recorded

in the eCRF as well as for data from other sources (e.g. laboratory).

13. TRIAL COMMITTEES

13.1. Clinical Events Committee

An independent Clinical Events Committee (CEC) will be established. The CEC will consist of

physicians who have no affiliation with the CardioMEMS<sup>TM</sup> HF System trial, are not employees


of Abbott Laboratories, or have no significant investment in Abbott Laboratories or their entities.

This committee will be composed of at least 3 members from which at least two are HF

cardiologists. Events for adjudication will include primary endpoints and device or procedure

related adverse events. Criteria for adjudication, procedures, data flow will be described in separate

CEC charter generated and maintained by the MHICC.

13.2. Data and Safety Monitoring Board (DSMB)

An independent Data and Safety Monitoring Board (DSMB) will be established. The DSMB is

responsible for safeguarding the interests of study participants, assessing the safety of study

procedures and for monitoring the overall conduct of the study The DSMB will consist of three

experienced physicians with expertise in clinical trial conduct. The DSMB will meet by

teleconference once a year, with additional meetings or conference calls scheduled as needed.


## **Proposed Table 1. Patient Characteristics at Enrollment**

| | Standard care | Virtual clinic | p value |
|---|---|---|---|
| Demographics and clinical | | | |
| Age, | | | |
| Gender | | | |
| Weight | | | |
| Body Mass Index (BMI) | | | |
| NYHA class, median (range) | | | |
| Heart rate, bpm | | | |
| Systolic blood pressure, mmHg | | | |
| Diastolic blood pressure, mmHg | | | |
| Medical History | | | |
| Dyslipidemia, % | | | |
| Diabetes mellitus, % | | | |
| Hypertension, % | | | |
| Aetiology of HF, % ischemic | | | |
| Prior myocardial infarction, % | | | |
| CABG, % | | | |
| Percutaneous coronary intervention, | | | |
| % | | | |
| Stroke | | | |
| Atrial fibrillation, % | | | |
| Sustained Ventricular Arrhythmias, % | | | |
| CRT, % | | | |
| ICD, % | | | |
| Pacemaker, % | | | |
| <u>Medications</u> | | | |
| ACEi/ARB, % | | | |
| ARNi, % | | | |
| B-blockers, % | | | |
| MRA, % | | | |
| Ivabradine, % | | | |
| Digoxin, % | | | |
| Hydralazine/nitrates, % | | | |
| Loop diuretics, % | | | |
| Other diuretics, % | | | |
| <u>Laboratory testing</u> <sup>#</sup> | | | |
| Sodium, mmol/l | | | |
| NT-proBNP, pg/mL | | | |
| BUN, mmol/L | | | |
| eGFR, mL/min/1.73 m2 (MDRD) | | | |
| Hemoglobin | | | |

| 6-Minute walk, m |
|-------------------------|
| Echocardiography# |
| LVEF, % |
| % with HFPEF (LVEF>40%) |
| LVESVI, ml |
| LAVi, ml |
| RV TAPSE |
| ePAPSP |
| PVR, Wood units |
| Resting hemodynamics& |
| RAP, mean, mm Hg |
| PAP, systolic, mm Hg |
| PAP, diastolic, mm Hg |
| PCWP, mm Hg |
| Cardiac output, L/min |
| Cardiac index, L/min/m2 |
| SVRI, dyne/ s/cm/m2 |
| PVR, Wood units |
| RVSWI, mL/beat/m2 |

<sup>#</sup> Selected parameters presented here; Data will likely be presented for HFrEF and HFpEF. & in implanted patients only.

NYHA indicates New York Heart Association; CRT, cardiac resynchronization therapy; ICD, implantable cardiac defibrillator; BNP, brain natriuretic peptide; eGFR, estimated glomerular filtration rate; LVEF, left ventricular ejection fraction; LVESVI: LV end systolic volume indexed to BSA; LAVi: Left atrial volume indexed to BSA; RV TAPSE: RV tricuspid annular plane systolic excursion, using Tissue Doppler imaging; eSPAP: estimated systolic PAP; PVR, pulmonary vascular resistance; RAP, right atrial pressure; PAP, pulmonary artery pressure; PCWP, pulmonary capillary wedge pressure; SVRI, systemic vascular resistance; and RVSWI, RV stroke work index.

Data will be summarized as mean±SD (range) unless otherwise specified.

## Proposed Table 2. Changes in the main Parameters between baseline and 12-months in Survivors

| | Standard care | Virtual clinic | p value |
|-------------------------------|---------------|----------------|---------|
| <u>Clinical</u> | | | |
| NYHA class, median (range) | | | |
| Heart rate, bpm | | | |
| Systolic blood pressure, mmHg | | | |
| 6-Minute walk, m | | | |
| MLHFQ | | | |
| Laboratory testing# | | | |
| Sodium, mmol/l | | | |
| NT-proBNP, pg/mL | | | |
| BUN, mmol/L | | | |
| eGFR, mL/min/1.73 m2 (MDRD) | | | |
| Hemoglobin | | | |
| Hs-CRP | | | |
| Troponin | | | |
| Osteopontin | | | |
| Angiotensin-2 | | | |
| Aldosterone | | | |
| Vasopressin | | | |
| PIIINP | | | |
| Galectin-3 | | | |
| ST2 | | | |
| Cystatin C | | | |
| Echocardiography <sup>#</sup> | | | |
| LVEF, % | | | |
| % with HFPEF (LVEF>40%) | | | |
| LVESVI, ml | | | |
| LAVi, ml | | | |
| RV TAPSE | | | |
| ePAPSP | | | |
| PVR, Wood units | | | |

<sup>\*</sup>Frailty index using the Fried scale<sup>40</sup>; # Selected parameters; final table will vary according to findings; & in implanted patients only.

NYHA indicates New York Heart Association; CRT, cardiac resynchronization therapy; ICD, implantable cardiac defibrillator; BNP, brain natriuretic peptide; eGFR, estimated glomerular filtration rate; LVEF, left ventricular ejection fraction; LVESVI: LV end systolic volume indexed to BSA; LAVi: Left atrial volume indexed to BSA; RV TAPSE: RV tricuspid annular plane systolic excursion, using Tissue Doppler imaging; eSPAP: estimated systolic PAP; PVR, pulmonary vascular resistance; RAP, right atrial pressure; PAP, pulmonary artery pressure; PCWP, pulmonary capillary wedge pressure; SVRI, systemic vascular resistance; and RVSWI, RV stroke work index. Data will be summarized as mean±SD (range) unless otherwise specified. p values will be for comparisons across all time points.


## Proposed Table 3. Pharmacological Profiles and Goal for best practice at 12 months

| | Standard care | | Virtual clinic | | p values | |
|---|---|---|---|---|---|---|
| MEDICATION | All | HFrEF | <u>HFpEF</u> | All | HFrEF | <b>HFpEF</b> |
| ACE or ARB, % and mean dose | | | | | | |
| % achieved target dose | | | NA | | | NA |
| ARNi, % and mean dose | | | | | | |
| % achieved target dose | | | | | | NA |
| β-blocker, % and mean dose | | | | | | |
| % achieved target dose | | | NA | | | NA |
| Mineralocorticoid receptors antagonist, % and mean dose | | | | | | |
| % achieved target dose | | | | | | |
| Ivabradine, % and mean dose | | | | | | |
| % achieved target dose | | | | | | |
| Loop diuretic, % and mean dose | | | | | | |
| Thiazide diuretic, % and mean dose | | | | | | |
| Digoxin, % and mean dose | | | | | | |
| Long-acting nitrates, % and mean dose | | | | | | |
| Hydralazine, % and mean dose | | | | | | |
| MEDICATION CHANGES | | | | | | |
| Number of medication changes/patient, mean, range | | | | | | |
| time (days) to achieve target doses of GDMT | | | | | | |

| * <i>P</i> for comparison between baseline and 12 months |
|----------------------------------------------------------|


## **Proposed Table 4: Device related endpoints**

- Safety: adverse events related to the device;
- number of successful patient contacts (virtual and clinic);
- PA pressures: changes, frequency of elevated readings


#### REFERENCES

- 1. Gheorghiade M, Zannad F, Sopko G, et al. Acute heart failure syndromes: current state and framework for future research. *Circulation*. 2005;112(25):3958-3968.
- 2. Fonarow GC, Abraham WT, Albert NM, et al. Association between performance measures and clinical outcomes for patients hospitalized with heart failure. *JAMA*. 2007;297(1):61-70.
- 3. Arnold JM, Howlett JG, Dorian P, et al. Canadian Cardiovascular Society Consensus Conference recommendations on heart failure update 2007: Prevention, management during intercurrent illness or acute decompensation, and use of biomarkers. *Can J Cardiol.* 2007;23(1):21-45.
- 4. Desai AS, Bhimaraj A, Bharmi R, et al. Ambulatory Hemodynamic Monitoring Reduces Heart Failure Hospitalizations in "Real-World" Clinical Practice. *J Am Coll Cardiol.* 2017;69(19):2357-2365.
- 5. Adamson PB. Pathophysiology of the transition from chronic compensated and acute decompensated heart failure: new insights from continuous monitoring devices. *Curr Heart Fail Rep.* 2009;6(4):287-292.
- 6. Simonneau G, Gatzoulis MA, Adatia I, et al. Updated clinical classification of pulmonary hypertension. *J Am Coll Cardiol*. 2013;62(25 Suppl):D34-D41.
- 7. Bursi F, McNallan SM, Redfield MM, et al. Pulmonary pressures and death in heart failure: a community study. *J Am Coll Cardiol*. 2012;59(3):222-231.
- 8. Ducharme A, Doyon O, White M, Rouleau JL, Brophy JM. Impact of care at a multidisciplinary congestive heart failure clinic: a randomized trial. *CMAJ.* 2005;173(1):40-45.
- 9. Ducharme A. Do Heart Failure Clinics Have to Reinvent Themselves to Remain Germane? *Can J Cardiol.* 2017;33(10):1212-1214.
- 10. Cleland JG, Louis AA, Rigby AS, Janssens U, Balk AH. Noninvasive home telemonitoring for patients with heart failure at high risk of recurrent admission and death: the Trans-European Network-Home-Care Management System (TEN-HMS) study. *J Am Coll Cardiol*. 2005;45(10):1654-1664.
- 11. Clark RA, Inglis SC, McAlister FA, Cleland JG, Stewart S. Telemonitoring or structured telephone support programmes for patients with chronic heart failure: systematic review and meta-analysis. *BMJ*. 2007;334(7600):942.
- 12. Chaudhry SI, Phillips CO, Stewart SS, et al. Telemonitoring for patients with chronic heart failure: a systematic review. *J Card Fail*. 2007;13(1):56-62.
- 13. Ong MK, Romano PS, Edgington S, et al. Effectiveness of Remote Patient Monitoring After Discharge of Hospitalized Patients With Heart Failure: The Better Effectiveness After Transition Heart Failure (BEAT-HF) Randomized Clinical Trial. *JAMA Intern Med.* 2016;176(3):310-318.
- 14. Morgan JM, Kitt S, Gill J, et al. Remote management of heart failure using implantable electronic devices. *Eur Heart J.* 2017.
- 15. Desai AS, Stevenson LW. Connecting the circle from home to heart-failure disease management. *N Engl J Med.* 2010;363(24):2364-2367.
- 16. van Veldhuisen DJ, Braunschweig F, Conraads V, et al. Intrathoracic impedance monitoring, audible patient alerts, and outcome in patients with heart failure. *Circulation*. 2011;124(16):1719-1726.


- 17. Boehmer JP, Hariharan R, Devecchi FG, et al. A Multisensor Algorithm Predicts Heart Failure Events in Patients With Implanted Devices: Results From the MultiSENSE Study. *JACC Heart Fail*. 2017:5(3):216-225.
- 18. Singh B, Russell SD, Cheng A. Update on device technologies for monitoring heart failure. *Curr Treat Options Cardiovasc Med.* 2012;14(5):536-549.
- 19. Adamson PB, Gold MR, Bennett T, et al. Continuous hemodynamic monitoring in patients with mild to moderate heart failure: results of The Reducing Decompensation Events Utilizing Intracardiac Pressures in Patients With Chronic Heart Failure (REDUCEhf) trial. *Congest Heart Fail.* 2011;17(5):248-254.
- 20. Ritzema J, Troughton R, Melton I, et al. Physician-directed patient self-management of left atrial pressure in advanced chronic heart failure. *Circulation*. 2010;121(9):1086-1095.
- 21. Troughton RW, Ritzema J, Eigler NL, et al. Direct left atrial pressure monitoring in severe heart failure: long-term sensor performance. *J Cardiovasc Transl Res.* 2011;4(1):3-13.
- 22. Maurer MS, Adamson PB, Costanzo MR, et al. Rationale and Design of the Left Atrial Pressure Monitoring to Optimize Heart Failure Therapy Study (LAPTOP-HF). *J Card Fail*. 2015;21(6):479-488.
- 23. William T.Abraham PBA, Maria Rosa Costanzo, Neal Eigler, Michaelold, Marc Klapholz, Mathew Maurer, Leslie Saxon, Jagmeet Singh, RichardTroughton. Hemodynamic Monitoring in Advanced Heart Failure: Results from the LAPTOP-HF Trial. *Journal of Cardiac Failure*. 2016;22(11):940.
- 24. Verdejo HE, Castro PF, Concepcion R, et al. Comparison of a radiofrequency-based wireless pressure sensor to swan-ganz catheter and echocardiography for ambulatory assessment of pulmonary artery pressure in heart failure. *J Am Coll Cardiol.* 2007;50(25):2375-2382.
- 25. Abraham WT, Adamson PB, Bourge RC, et al. Wireless pulmonary artery haemodynamic monitoring in chronic heart failure: a randomised controlled trial. *Lancet*. 2011;377(9766):658-666.
- 26. Benza RL, Raina A, Abraham WT, et al. Pulmonary hypertension related to left heart disease: insight from a wireless implantable hemodynamic monitor. *J Heart Lung Transplant*. 2015;34(3):329-337.
- 27. Adamson PB, Abraham WT, Bourge RC, et al. Wireless pulmonary artery pressure monitoring guides management to reduce decompensation in heart failure with preserved ejection fraction. *Circ Heart Fail.* 2014;7(6):935-944.
- 28. Fang JC, DeMarco T, Givertz MM, et al. World Health Organization Pulmonary Hypertension group 2: pulmonary hypertension due to left heart disease in the adult--a summary statement from the Pulmonary Hypertension Council of the International Society for Heart and Lung Transplantation. *J Heart Lung Transplant*. 2012;31(9):913-933.
- 29. Krahnke JS, Abraham WT, Adamson PB, et al. Heart failure and respiratory hospitalizations are reduced in patients with heart failure and chronic obstructive pulmonary disease with the use of an implantable pulmonary artery pressure monitoring device. *J Card Fail*. 2015;21(3):240-249.
- 30. Raina A, Abraham WT, Adamson PB, Bauman J, Benza RL. Limitations of right heart catheterization in the diagnosis and risk stratification of patients with pulmonary hypertension related to left heart disease: insights from a wireless pulmonary artery pressure monitoring system. *J Heart Lung Transplant*. 2015;34(3):438-447.
- 31. Binanay C, Califf RM, Hasselblad V, et al. Evaluation study of congestive heart failure and pulmonary artery catheterization effectiveness: the ESCAPE trial. *JAMA*. 2005;294(13):1625-1633.

- 32. Reiter MJ, Stromberg KD, Whitman TA, Adamson PB, Benditt DG, Gold MR. Influence of intracardiac pressure on spontaneous ventricular arrhythmias in patients with systolic heart failure: insights from the REDUCEhf trial. *Circ Arrhythm Electrophysiol.* 2013;6(2):272-278.
- 33. Ebinger MW, Krishnan S, Schuger CD. Mechanisms of ventricular arrhythmias in heart failure. *Curr Heart Fail Rep.* 2005;2(3):111-117.
- 34. Adamson PB, Smith AL, Abraham WT, et al. Continuous autonomic assessment in patients with symptomatic heart failure: prognostic value of heart rate variability measured by an implanted cardiac resynchronization device. *Circulation*. 2004;110(16):2389-2394.
- 35. Reiter MJ. Effects of mechano-electrical feedback: potential arrhythmogenic influence in patients with congestive heart failure. *Cardiovasc Res.* 1996;32(1):44-51.
- 36. Schmier JK, Ong KL, Fonarow GC. Cost-Effectiveness of Remote Cardiac Monitoring With the CardioMEMS Heart Failure System. *Clin Cardiol*. 2017;40(7):430-436.
- 37. Adamson PB, Abraham WT, Stevenson LW, et al. Pulmonary Artery Pressure-Guided Heart Failure Management Reduces 30-Day Readmissions. *Circ Heart Fail.* 2016;9(6).
- 38. Nerenberg KA, Zarnke KB, Leung AA, et al. Hypertension Canada's 2018 Guidelines for Diagnosis, Risk Assessment, Prevention, and Treatment of Hypertension in Adults and Children. *Can J Cardiol.* 2018;34(5):506-525.
- 39. Levey AS, Bosch JP, Lewis JB, Greene T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation. Modification of Diet in Renal Disease Study Group. *Ann Intern Med.* 1999;130(6):461-470.
- 40. Iwanaga Y, Miyazaki S. Heart failure, chronic kidney disease, and biomarkers--an integrated viewpoint. *Circ J.* 74(7):1274-1282.
- 41. de Denus S, Pharand C, Williamson DR. Brain natriuretic peptide in the management of heart failure: the versatile neurohormone. *Chest.* 2004;125(2):652-668.
- 42. Skaf S, Thibault B, Khairy P, et al. Impact of Left Ventricular vs Biventricular Pacing on Reverse Remodelling: Insights From the Evaluation of Resynchronization Therapy for Heart Failure (EARTH) Trial. *Can J Cardiol.* 2017;33(10):1274-1282.
- 43. Thibault B, Ducharme A, Harel F, et al. Left ventricular versus simultaneous biventricular pacing in patients with heart failure and a QRS complex >/=120 milliseconds. *Circulation*. 2011;124(25):2874-2881.
- 44. White M, Lepage S, Lavoie J, et al. Effects of combined candesartan and ACE inhibitors on BNP, markers of inflammation and oxidative stress, and glucose regulation in patients with symptomatic heart failure. *J Card Fail.* 2007;13(2):86-94.
- de Denus S, Lavoic J, Ducharme A, et al. Differences in concentrations and correlations amongst biomarkers of neurohormonal activation, inflammation and extracellular matrix turnover in patients with HF and a reduced or a preserved left ventricular ejection fraction. *Journal of Cardiac Failure*. 2008;14(6):S38-S38.
- 46. Lopez B, Gonzalez A, Varo N, Laviades C, Querejeta R, Diez J. Biochemical assessment of myocardial fibrosis in hypertensive heart disease. *Hypertension*. 2001;38(5):1222-1226.
- 47. Nishikawa N, Yamamoto K, Sakata Y, et al. Differential activation of matrix metalloproteinases in heart failure with and without ventricular dilatation. *Cardiovasc Res.* 2003;57(3):766-774.


48. Zannad F, Radauceanu A. Effect of MR blockade on collagen formation and cardiovascular disease with a specific emphasis on heart failure. *Heart Fail Rev.* 2005;10(1):71-78.

- 49. Cicoira M, Rossi A, Bonapace S, et al. Independent and additional prognostic value of aminoterminal propeptide of type III procollagen circulating levels in patients with chronic heart failure. *J Card Fail.* 2004;10(5):403-411.
- 50. Zannad F, Alla F, Dousset B, Perez A, Pitt B. Limitation of excessive extracellular matrix turnover may contribute to survival benefit of spironolactone therapy in patients with congestive heart failure: insights from the randomized aldactone evaluation study (RALES). Rales Investigators. *Circulation*. 2000;102(22):2700-2706.
- 51. Tsutamoto T, Wada A, Maeda K, et al. Effect of spironolactone on plasma brain natriuretic peptide and left ventricular remodeling in patients with congestive heart failure. *J Am Coll Cardiol*. 2001;37(5):1228-1233.
- 52. Macdonald JE, Kennedy N, Struthers AD. Effects of spironolactone on endothelial function, vascular angiotensin converting enzyme activity, and other prognostic markers in patients with mild heart failure already taking optimal treatment. *Heart*. 2004;90(7):765-770.
- O'Meara E, Rouleau JL, White M, et al. Heart failure with anemia: novel findings on the roles of renal disease, interleukins, and specific left ventricular remodeling processes. *Circ Heart Fail*. 2014;7(5):773-781.
- 54. Spinale FG. Myocardial matrix remodeling and the matrix metalloproteinases: influence on cardiac form and function. *Physiol Rev.* 2007;87(4):1285-1342.
- Ashkar S, Glimcher MJ, Saavedra RA. Mouse osteopontin expressed in E. coli exhibits autophosphorylating activity of tyrosine residues. *Biochem Biophys Res Commun.* 1993;194(1):274-279.
- 56. Ashkar S, Weber GF, Panoutsakopoulou V, et al. Eta-1 (osteopontin): an early component of type-1 (cell-mediated) immunity. *Science*. 2000;287(5454):860-864.
- 57. Iraqi W, Rossignol P, Angioi M, et al. Extracellular cardiac matrix biomarkers in patients with acute myocardial infarction complicated by left ventricular dysfunction and heart failure: insights from the Eplerenone Post-Acute Myocardial Infarction Heart Failure Efficacy and Survival Study (EPHESUS) study. *Circulation*. 2009;119(18):2471-2479.
- 58. Ahmad T, Fiuzat M, Neely B, et al. Biomarkers of myocardial stress and fibrosis as predictors of mode of death in patients with chronic heart failure. *JACC Heart Fail*. 2014;2(3):260-268.
- 59. Chaikijurajai T, Tang WHW. Reappraisal of Inflammatory Biomarkers in Heart Failure. *Curr Heart Fail Rep.* 2020.
- 60. Meijers WC, Januzzi JL, deFilippi C, et al. Elevated plasma galectin-3 is associated with near-term rehospitalization in heart failure: a pooled analysis of 3 clinical trials. *Am Heart J.* 2014;167(6):853-860 e854.
- 61. Shah RV, Chen-Tournoux AA, Picard MH, van Kimmenade RR, Januzzi JL. Galectin-3, cardiac structure and function, and long-term mortality in patients with acutely decompensated heart failure. *Eur J Heart Fail.* 2010;12(8):826-832.
- 62. Shah RV, Januzzi JL, Jr. Soluble ST2 and galectin-3 in heart failure. *Clin Lab Med.* 2014;34(1):87-97, vi-vii.
- 63. Zilinski JL, Shah RV, Gaggin HK, Gantzer ML, Wang TJ, Januzzi JL. Measurement of multiple biomarkers in advanced stage heart failure patients treated with pulmonary artery catheter guided therapy. *Crit Care*. 2012;16(4):R135.
- 64. Simpson CE, Damico RL, Hassoun PM, et al. Noninvasive prognostic biomarkers for left heart failure as predictors of survival in pulmonary arterial hypertension. *Chest.* 2020.

Protocol No: MHICC-2018-001 Version: FINAL 10

- 65. Lubrano V, Balzan S. Role of oxidative stress-related biomarkers in heart failure: galectin 3, alpha1-antitrypsin and LOX-1: new therapeutic perspective? *Mol Cell Biochem.* 2020;464(1-2):143-152.
- 66. She G, Hou MC, Zhang Y, et al. Gal-3 (Galectin-3) and KCa3.1 Mediate Heterogeneous Cell Coupling and Myocardial Fibrogenesis Driven by betaAR (beta-Adrenoceptor) Activation. *Hypertension*. 2020;75(2):393-404.
- 67. Shah RV, Chen-Tournoux AA, Picard MH, van Kimmenade RR, Januzzi JL. Serum levels of the interleukin-1 receptor family member ST2, cardiac structure and function, and long-term mortality in patients with acute dyspnea. *Circ Heart Fail*. 2009;2(4):311-319.
- 68. Shah RV, Januzzi JL, Jr. ST2: a novel remodeling biomarker in acute and chronic heart failure. *Curr Heart Fail Rep.* 2010;7(1):9-14.
- 69. Iovino M, Iacoviello M, De Pergola G, et al. Vasopressin in Heart Failure. *Endocr Metab Immune Disord Drug Targets*. 2018;18(5):458-465.
- 70. Chirinos JA, Sardana M, Oldland G, et al. Association of arginine vasopressin with low atrial natriuretic peptide levels, left ventricular remodelling, and outcomes in adults with and without heart failure. *ESC Heart Fail*. 2018;5(5):911-919.
- 71. Ogawa R, Stachnik JM, Echizen H. Clinical pharmacokinetics of drugs in patients with heart failure: an update (part 2, drugs administered orally). *Clin Pharmacokinet*. 2014;53(12):1083-1114.
- 72. Gonzalez O, Alonso RM, Ferreirós N, Weinmann W, Zimmermann R, Dresen S. Development of an LC–MS/MS method for the quantitation of 55 compounds prescribed in combined cardiovascular therapy. *Journal of Chromatography B*. 2011;879(3):243-252.
- 73. Gundersen POM, Helland A, Spigset O, Hegstad S. Quantification of 21 antihypertensive drugs in serum using UHPLC-MS/MS. *Journal of Chromatography B*. 2018;1089:84-93.
- 74. Dias E, Hachey B, McNaughton C, et al. An LC–MS assay for the screening of cardiovascular medications in human samples. *Journal of Chromatography B.* 2013;937:44-53.
- 75. Gonzalez O, Iriarte G, Rico E, et al. LC–MS/MS method for the determination of several drugs used in combined cardiovascular therapy in human plasma. *Journal of Chromatography B.* 2010;878(28):2685-2692.
- 76. De Nicolò A, Avataneo V, Rabbia F, et al. UHPLC–MS/MS method with protein precipitation extraction for the simultaneous quantification of ten antihypertensive drugs in human plasma from resistant hypertensive patients. *Journal of Pharmaceutical and Biomedical Analysis*. 2016;129:535-541.
- 77. Joye T, Sidibé J, Déglon J, et al. Liquid chromatography-high resolution mass spectrometry for broad-spectrum drug screening of dried blood spot as microsampling procedure. *Analytica Chimica Acta*. 2019;1063:110-116.
- 78. Rosano TG, Ohouo PY, Wood M. Application of High-Resolution UPLC–MSE/TOF Confirmation in Forensic Urine Drug Screening by UPLC–MS/MS. *Journal of Analytical Toxicology*. 2019;43(5):353-363.
- 79. Mollerup CB, Dalsgaard PW, Mardal M, Linnet K. Targeted and non-targeted drug screening in whole blood by UHPLC-TOF-MS with data-independent acquisition. *Drug Testing and Analysis*. 2017;9(7):1052-1061.
- 80. Kim EH, Seo HS, Ki NY, et al. Reliable screening and confirmation of 156 multi-class illegal adulterants in dietary supplements based on extracted common ion chromatograms by ultrahigh-performance liquid chromatography-quadrupole/time of flight-mass spectrometry. *Journal of Chromatography A*. 2017;1491:43-56.

- 81. Richter LHJ, Jacobs CM, Mahfoud F, Kindermann I, Böhm M, Meyer MR. Development and application of a LC-HRMS/MS method for analyzing antihypertensive drugs in oral fluid for monitoring drug adherence. *Analytica Chimica Acta*. 2019;1070:69-79.
- 82. Tomková J, Ondra P, Kocianová E, Václavík J. Fast and sensitive analysis of beta blockers by ultra-high-performance liquid chromatography coupled with ultra-high-resolution TOF mass spectrometry. *Biomedical Chromatography*. 2017;31(7):e3911.
- 83. Hossain MA, Friciu M, Aubin S, Leclair G. Stability of penicillin G sodium diluted with 0.9% sodium chloride injection or 5% dextrose injection and stored in polyvinyl chloride bag containers and elastomeric pump containers. *Am J Health Syst Pharm.* 2014;71(8):669-673.
- 84. Li M, Coursol C, Leclair G. Stability of cyclosporine diluted with 0.9% sodium chloride injection or 5% dextrose injection and stored in ethylene-vinyl acetate containers. *Am J Health Syst Pharm*. 2013;70(22):1970-1972.
- 85. Li M, Forest JM, Coursol C, Leclair G. Stability of cyclosporine solutions stored in polypropylene-polyolefin bags and polypropylene syringes. *Am J Health Syst Pharm.* 2011;68(17):1646-1650.
- 86. Friciu M, Chefson A, Leclair G. Stability of Hydrocortisone, Nifedipine, and Nitroglycerine Compounded Preparations for the Treatment of Anorectal Conditions. *Can J Hosp Pharm.* 2016;69(4):329-333.
- 87. Friciu M, Zaraa S, Leclair G. Stability of Extemporaneously Prepared Enalapril Maleate Suspensions in Glass Bottles and Plastic Syringes. *Can J Hosp Pharm.* 2016;69(6):505-507.
- 88. Friciu M, Zaraa S, Leclair G. Stability of Extemporaneously Compounded Amlodipine Besylate Oral Suspensions. *Can J Hosp Pharm.* 2016;69(4):327-329.
- 89. Friciu M, Zaraa S, Leclair G. Stability of Extemporaneously Compounded Tacrolimus in Glass Bottles and Plastic Syringes. *Can J Hosp Pharm.* 2017;70(1):51-53.
- 90. Sullivan T, Forest JM, Leclair G. Compatibility of Cloxacillin Sodium with Selected Intravenous Drugs During Simulated Y-Site Administration. *Hosp Pharm.* 2015;50(3):214-220.
- 91. Friciu M, Plourde K, Leclair G, Danopoulos P, Savji T. Stability of Prednisone in Oral Mix Suspending Vehicle. *Int J Pharm Compd.* 2015;19(4):337-339.
- 92. Melkoumov A, Goupil M, Louhichi F, Raymond M, de Repentigny L, Leclair G. Nystatin nanosizing enhances in vitro and in vivo antifungal activity against Candida albicans. *J Antimicrob Chemother*. 2013;68(9):2099-2105.
- 93. Friciu M, Roullin VG, Leclair G. Stability of gabapentin in extemporaneously compounded oral suspensions. *PLoS One.* 2017;12(4):e0175208.
- 94. Friciu M, Zaraa S, Roullin VG, Leclair G. Stability of Diazoxide in Extemporaneously Compounded Oral Suspensions. *PLoS One.* 2016;11(10):e0164577.
- 95. Korol S, White M, O'Meara E, et al. A comparison of the effects of selective and non-selective mineralocorticoid antagonism on glucose homeostasis of heart failure patients with glucose intolerance or type II diabetes: A randomized controlled double-blind trial. *Am Heart J.* 2018;204:190-195.
- 96. Collin-Levesque L, El-Ghaddaf Y, Genest M, et al. Infant Exposure to Methylphenidate and Duloxetine During Lactation. *Breastfeed Med.* 2018;13(3):221-225.
- 97. de Denus S, O'Meara E, Desai AS, et al. Spironolactone Metabolites in TOPCAT New Insights into Regional Variation. *N Engl J Med.* 2017;376(17):1690-1692.
- 98. Sheiner LB, Rosenberg B, Melmon KL. Modelling of individual pharmacokinetics for computer-aided drug dosage. *Comput Biomed Res.* 1972;5(5):411-459.
- 99. Mould DR, Upton RN. Basic concepts in population modeling, simulation, and model-based drug development. *CPT Pharmacometrics Syst Pharmacol.* 2012;1:e6.

- 100. Marsot A, Boulamery A, Bruguerolle B, Simon N. Vancomycin: a review of population pharmacokinetic analyses. *Clin Pharmacokinet*. 2012;51(1):1-13.
- 101. Marsot A, Brevaut-Malaty V, Vialet R, Boulamery A, Bruguerolle B, Simon N. Pharmacokinetics and absolute bioavailability of phenobarbital in neonates and young infants, a population pharmacokinetic modelling approach. *Fundam Clin Pharmacol.* 2014;28(4):465-471.
- 102. Marsot A, Gallais F, Galambrun C, et al. Vancomycin in Pediatric Patients with Solid or Hematological Malignant Disease: Predictive Performance of a Population Pharmacokinetic Model and New Optimized Dosing Regimens. *Paediatr Drugs.* 2018;20(4):375-381.
- 103. Marsot A, Guilhaumou R, Riff C, Blin O. Amikacin in Critically III Patients: A Review of Population Pharmacokinetic Studies. *Clin Pharmacokinet*. 2017;56(2):127-138.
- 104. Marsot A, Imbert B, Alvarez JC, et al. High variability in the exposure of baclofen in alcohol-dependent patients. *Alcohol Clin Exp Res.* 2014;38(2):316-321.
- 105. Marsot A, Menard A, Dupouey J, Muziotti C, Guilhaumou R, Blin O. Population pharmacokinetics of rifampicin in adult patients with osteoarticular infections: interaction with fusidic acid. *Br J Clin Pharmacol.* 2017;83(5):1039-1047.
- 106. Marsot A, Michel F, Chasseloup E, Paut O, Guilhaumou R, Blin O. Phenobarbital in intensive care unit pediatric population: predictive performances of population pharmacokinetic model. *Fundam Clin Pharmacol.* 2017;31(5):558-566.
- 107. Marsot A, Vialet R, Boulamery A, Bruguerolle B, Simon N. Vancomycin: Predictive Performance of a Population Pharmacokinetic Model and Optimal Dose in Neonates and Young Infants. *Clin Pharmacol Drug Dev.* 2012;1(4):144-151.
- 108. Thirion DJG, Pasche V, Marsot A. What is the recommended amikacin dosing for cystic fibrosis patients with acute pulmonary exacerbations? *Pediatr Pulmonol.* 2019;54(11):1652-1653.

**Appendix 1: Elevated PA Mean Pressure – General Treatment Strategies in Protocol** 



Ultimate treatment decisions to be made by the Investigator

\*Minimum weekly review of PA mean trends


# Appendix 2: Hospital admissions at Montreal Heart Institute with a primary diagnosis of heart failure, financial year April 1st 2016 to March 31st 2017

### Heart Failure

APRIL 1st 2018 TO MARCH 31st 2019

| #<br>hospitalizations | # Pts | Mean age | men | women | # emergency<br>department<br>consultations |
|---|---|---|---|---|---|
| 900 | 716 | 76 | 281 | 435 | 1393 |

39,20% 60,80%

| Nb Readmission during the same financial year * | |
|-------------------------------------------------|-------|
| # Readmission | # pts |
| 0 | 475 |
| 1 | 135 |
| 2 | 65 |
| 3 | 32 |
| 4 | 5 |
| 5 | 2 |
| 6 | 1 |
| 7 | 0 |
| 8 | 0 |
| 9 | 1 |

716

Source: Karine Pearson, MHI archives, September 23, 2019


<sup>\*</sup> nb of readmission after a first HF episode

## Appendix 3: Example of an individualized therapeutic plan

#### Hypovolemic

PASP < 15 mmHg

PADP < 8 PAM < 25

#### Optivolemic

PASP 15-35 mmHg

PADP 8-20 PAM 10-25

#### Elevated PAP

PASP > 35 mmHg"

PADP > 20

PAM > 25

Reduced PAP:

Dehydratation, overdiuresis

Elevated PAP:

Volume overload, PH, ischemia, MR,

Persistent PH

Hold/reduce diuretics

Avoid reducing ARE/ARB, β-blockers unless no other options

Advance

ACE/ARB,

β-blockers and

MRA

to Target/tolerance

Advance ACE/ARB, β-blockers and MRA to Target/tolerance

Consider adding

hydralazine– nitrates

digoxin

RANGE PADP: low 5-8 Very low 0-5 optimal: 8-20 High: 20 -30 Very high > 30 AM Loop Diuretic hold 1/2 dose no change X 1.5 dose X 2 dose PM nitrates hold 1/2 dose no change X 1.5 dose X 2 dose hold fluid restriction X 24H ? dietary restriction Call nurse if symptoms instructions: (fluid & Na+)

Clinic or remote follow-up more frequently

Or PRN if symptoms

Control labs 1 week

As per protocol

PRN if symptoms

Clinic or remote follow-up more frequently

Or PRN if symptoms

Control labs 1 week

Modified from: MS Maurer et al. J Cardiac Failure 2015 and WT Abraham et al. Lancet 2011


**Clinical Review & Education** 

#### Special Communication

## World Medical Association Declaration of Helsinki Ethical Principles for Medical Research Involving Human Subjects

World Medical Association

Adopted by the 18th WMA General Assembly, Helsinki, Finland, June 1964, and amended by the:
29th WMA General Assembly, Tokyo, Japan, October 1975
35th WMA General Assembly, Venice, Italy, October 1983
41st WMA General Assembly, Hong Kong, September 1989
48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996
52nd WMA General Assembly, Edinburgh, Scotland, October 2000
53rd WMA General Assembly, Washington, DC, USA, October 2002 (Note of Clarification added)
55th WMA General Assembly, Tokyo, Japan, October 2004 (Note of Clarification added)
59th WMA General Assembly, Seoul, Republic of Korea, October 2008
64th WMA General Assembly, Fortaleza, Brazil, October 2013

#### Preamble

 The World Medical Association (WMA) has developed the Declaration of Helsinki as a statement of ethical principles for medical research involving human subjects, including research on identifiable human material and data.

The Declaration is intended to be read as a whole and each of its constituent paragraphs should be applied with consideration of all other relevant paragraphs.

Consistent with the mandate of the WMA, the Declaration is addressed primarily to physicians. The WMA encourages others who are involved in medical research involving human subjects to adopt these principles.

#### **General Principles**

- The Declaration of Geneva of the WMA binds the physician with the words, "The health of my patient will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act in the patient's best interest when providing medical care."
- 4. It is the duty of the physician to promote and safeguard the health, well-being and rights of patients, including those who are involved in medical research. The physician's knowledge and conscience are dedicated to the fulfilment of this duty.
- Medical progress is based on research that ultimately must include studies involving human subjects.
- The primary purpose of medical research involving human subjects is to understand the causes, development and effects of diseases and improve preventive, diagnostic and therapeutic interventions (methods, procedures and treatments). Even the

best proven interventions must be evaluated continually through research for their safety, effectiveness, efficiency, accessibility and quality.

- Medical research is subject to ethical standards that promote and ensure respect for all human subjects and protect their health and rights.
- While the primary purpose of medical research is to generate new knowledge, this goal can never take precedence over the rights and interests of individual research subjects.
- 9. It is the duty of physicians who are involved in medical research to protect the life, health, dignity, integrity, right to selfdetermination, privacy, and confidentiality of personal information of research subjects. The responsibility for the protection of research subjects must always rest with the physician or other health care professionals and never with the research subjects, even though they have given consent.
- 10. Physicians must consider the ethical, legal and regulatory norms and standards for research involving human subjects in their own countries as well as applicable international norms and standards. No national or international ethical, legal or regulatory requirement should reduce or eliminate any of the protections for research subjects set forth in this Declaration.
- Medical research should be conducted in a manner that minimises possible harm to the environment.
- 12. Medical research involving human subjects must be conducted only by individuals with the appropriate ethics and scientific education, training and qualifications. Research on patients or healthy volunteers requires the supervision of a competent and appropriately qualified physician or other health care professional.

2191

JAMA November 27, 2013 Volume 310, Number 20

- Groups that are underrepresented in medical research should be provided appropriate access to participation in research.
- 14. Physicians who combine medical research with medical care should involve their patients in research only to the extent that this is justified by its potential preventive, diagnostic or therapeutic value and if the physician has good reason to believe that participation in the research study will not adversely affect the health of the patients who serve as research subjects.
- Appropriate compensation and treatment for subjects who are harmed as a result of participating in research must be ensured.

#### Risks, Burdens and Benefits

 In medical practice and in medical research, most interventions involve risks and burdens.

Medical research involving human subjects may only be conducted if the importance of the objective outweighs the risks and burdens to the research subjects.

17. All medical research involving human subjects must be preceded by careful assessment of predictable risks and burdens to the individuals and groups involved in the research in comparison with foreseeable benefits to them and to other individuals or groups affected by the condition under investigation.

Measures to minimise the risks must be implemented. The risks must be continuously monitored, assessed and documented by the researcher.

 Physicians may not be involved in a research study involving human subjects unless they are confident that the risks have been adequately assessed and can be satisfactorily managed.

When the risks are found to outweigh the potential benefits or when there is conclusive proof of definitive outcomes, physicians must assess whether to continue, modify or immediately stop the study.

#### Vulnerable Groups and Individuals

 Some groups and individuals are particularly vulnerable and may have an increased likelihood of being wronged or of incurring additional harm.

All vulnerable groups and individuals should receive specifically considered protection.

20. Medical research with a vulnerable group is only justified if the research is responsive to the health needs or priorities of this group and the research cannot be carried out in a nonvulnerable group. In addition, this group should stand to benefit from the knowledge, practices or interventions that result from the research.

#### Scientific Requirements and Research Protocols

- Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and adequate laboratory and, as appropriate, animal experimentation. The welfare of animals used for research must be respected.
- The design and performance of each research study involving human subjects must be clearly described and justified in a research protocol.

The protocol should contain a statement of the ethical considerations involved and should indicate how the principles in this Declaration have been addressed. The protocol should include information regarding funding, sponsors, institutional affiliations, potential conflicts of interest, incentives for subjects and information regarding provisions for treating and/or compensating subjects who are harmed as a consequence of participation in the research study.

In clinical trials, the protocol must also describe appropriate arrangements for post-trial provisions.

#### Research Ethics Committees

23. The research protocol must be submitted for consideration, comment, guidance and approval to the concerned research ethics committee before the study begins. This committee must be transparent in its functioning, must be independent of the researcher, the sponsor and any other undue influence and must be duly qualified. It must take into consideration the laws and regulations of the country or countries in which the research is to be performed as well as applicable international norms and standards but these must not be allowed to reduce or eliminate any of the protections for research subjects set forth in this Declaration.

The committee must have the right to monitor ongoing studies. The researcher must provide monitoring information to the committee, especially information about any serious adverse events. No amendment to the protocol may be made without consideration and approval by the committee. After the end of the study, the researchers must submit a final report to the committee containing a summary of the study's findings and conclusions.

#### **Privacy and Confidentiality**

 Every precaution must be taken to protect the privacy of research subjects and the confidentiality of their personal information.

#### Informed Consent

 Participation by individuals capable of giving informed consent as subjects in medical research must be voluntary. Although it

192 JAMA November 27, 2013 Volume 310, Number 20

Jama.com

Copyright 2013 American Medical Association. All rights reserved.

Protocol No: MHICC-2018-001 Version: FINAL 10

may be appropriate to consult family members or community leaders, no individual capable of giving informed consent may be enrolled in a research study unless he or she freely agrees.

26. In medical research involving human subjects capable of giving informed consent, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail, post-study provisions and any other relevant aspects of the study. The potential subject must be informed of the right to refuse to participate in the study or to withdraw consent to participate at any time without reprisal. Special attention should be given to the specific information needs of individual potential subjects as well as to the methods used to deliver the information.

After ensuring that the potential subject has understood the information, the physician or another appropriately qualified individual must then seek the potential subject's freely-given informed consent, preferably in writing. If the consent cannot be expressed in writing, the non-written consent must be formally documented and witnessed.

All medical research subjects should be given the option of being informed about the general outcome and results of the study.

- 27. When seeking informed consent for participation in a research study the physician must be particularly cautious if the potential subject is in a dependent relationship with the physician or may consent under duress. In such situations the informed consent must be sought by an appropriately qualified individual who is completely independent of this relationship.
- 28. For a potential research subject who is incapable of giving informed consent, the physician must seek informed consent from the legally authorised representative. These individuals must not be included in a research study that has no likelihood of benefit for them unless it is intended to promote the health of the group represented by the potential subject, the research cannot instead be performed with persons capable of providing informed consent, and the research entails only minimal risk and minimal burden.
- 29. When a potential research subject who is deemed incapable of giving informed consent is able to give assent to decisions about participation in research, the physician must seek that assent in addition to the consent of the legally authorised representative. The potential subject's dissent should be respected.
- 30. Research involving subjects who are physically or mentally incapable of giving consent, for example, unconscious patients, may be done only if the physical or mental condition that prevents giving informed consent is a necessary characteristic of the research group. In such circumstances the physician must seek informed consent from the legally authorised representative. If no such representative is available and if the research cannot be delayed, the study may proceed without informed consent pro-

vided that the specific reasons for involving subjects with a condition that renders them unable to give informed consent have been stated in the research protocol and the study has been approved by a research ethics committee. Consent to remain in the research must be obtained as soon as possible from the subject or a legally authorised representative.

- 31. The physician must fully inform the patient which aspects of their care are related to the research. The refusal of a patient to participate in a study or the patient's decision to withdraw from the study must never adversely affect the patient-physician relationship.
- 32. For medical research using identifiable human material or data, such as research on material or data contained in biobanks or similar repositories, physicians must seek informed consent for its collection, storage and/or reuse. There may be exceptional situations where consent would be impossible or impracticable to obtain for such research. In such situations the research may be done only after consideration and approval of a research ethics committee.

#### Use of Placebo

33. The benefits, risks, burdens and effectiveness of a new intervention must be tested against those of the best proven intervention(s), except in the following circumstances:

Where no proven intervention exists, the use of placebo, or no intervention, is acceptable; or

Where for compelling and scientifically sound methodological reasons the use of any intervention less effective than the best proven one, the use of placebo, or no intervention is necessary to determine the efficacy or safety of an intervention

and the patients who receive any intervention less effective than the best proven one, placebo, or no intervention will not be subject to additional risks of serious or irreversible harm as a result of not receiving the best proven intervention.

Extreme care must be taken to avoid abuse of this option.

#### Post-Trial Provisions

34. In advance of a clinical trial, sponsors, researchers and host country governments should make provisions for post-trial access for all participants who still need an intervention identified as beneficial in the trial. This information must also be disclosed to participants during the informed consent process.

## Research Registration and Publication and Dissemination of Results

 Every research study involving human subjects must be registered in a publicly accessible database before recruitment of the first subject.

jama.com

JAMA November 27, 2013 Volume 310, Number 20 2193

Copyright 2013 American Medical Association. All rights reserved.

Protocol No: MHICC-2018-001 Version: FINAL 10

36. Researchers, authors, sponsors, editors and publishers all have ethical obligations with regard to the publication and dissemination of the results of research. Researchers have a duty to make publicly available the results of their research on human subjects and are accountable for the completeness and accuracy of their reports. All parties should adhere to accepted guidelines for ethical reporting. Negative and inconclusive as well as positive results must be published or otherwise made publicly available. Sources of funding, institutional affiliations and conflicts of interest must be declared in the publication. Reports of research not in accordance with the principles of this Declaration should not be accepted for publication.

#### Unproven Interventions in Clinical Practice

37. In the treatment of an individual patient, where proven interventions do not exist or other known interventions have been ineffective, the physician, after seeking expert advice, with informed consent from the patient or a legally authorised representative, may use an unproven intervention if in the physician's judgement it offers hope of saving life, re-establishing health or alleviating suffering. This intervention should subsequently be made the object of research, designed to evaluate its safety and efficacy. In all cases, new information must be recorded and, where appropriate, made publicly available.

#### ARTICLE INFORMATION

Corresponding Author: World Medical Association, 13, ch. du Levant, CIB - Bâtiment A, 01210 Ferney-Voltaire, France; wma@wma.net. Published Online: October 19, 2013. dol:10.1001/jama.2013.281053. Disclaimer: ©2013 World Medical Association, Inc. All Rights Reserved. All intellectual property rights in the Declaration of Helsinki are vested in the World Medical Association. The WMA has granted JAMA exclusive rights to publish the English-language version of the Declaration through December 31, 2013.

Online-Only Content: Audio podcast is available at www.lama.com.

Protocol No: MHICC-2018-001 Version: FINAL 10